J2T-MC-KGBO: Statistical Analysis Plan Version 2

An Open-Label Study to Evaluate the Safety and Efficacy of Lebrikizumab in Adult and Adolescent Participants with Moderate-to-Severe Atopic Dermatitis Previously Treated with Dupilumab

NCT05369403

Approval Date: 23-Jun-2023

# **Statistical Analysis Plan:**

J2T-MC-KGBO (Lebrikizumab): An Open-Label Study to Evaluate the Safety and Efficacy of Lebrikizumab in Adult and Adolescent Participants with Moderate-to-Severe Atopic Dermatitis Previously Treated with Dupilumab

### **Confidential Information**

The information contained in this document is confidential and the information contained within it may not be reproduced or otherwise disseminated without the approval of Eli Lilly and Company or its subsidiaries.

Note to Regulatory Authorities: This document may contain protected personal data and/or commercially confidential information exempt from public disclosure. Eli Lilly and Company requests consultation regarding release/redaction prior to any public release. In the United States, this document is subject to Freedom of Information Act (FOIA) Exemption 4 and may not be reproduced or otherwise disseminated without the written approval of Eli Lilly and Company or its subsidiaries.

Lebrikizumab (LY3650150)

Eli Lilly and Company Indianapolis, Indiana USA 46285 [Protocol J2T-MC-KGBO] [Phase 3b]

Statistical Analysis Plan Version 2

# **1.Table of Contents**

| Section | Page |
|--------------------------------------------------------------|------|
| 1. Table of Contents | 2 |
| 2. Revision History | 8 |
| 3. Study Objectives | 9 |
| 4. Study Design | |
| 4.1. Summary of Study Design | |
| 4.1.1 Number of Participants | |
| 4.1.2 Schema | |
| 4.2. Determination of Sample Size | |
| 4.3. Method of Assignment to Treatment | |
| 5. A Priori Statistical Methods | 14 |
| 5.1. General Considerations | |
| 5.1.1. Analysis Populations | |
| 5.1.2. General Considerations for Analyses | |
| 5.2. Primary and Supportive Estimands | |
| 5.2.1. Primary Estimand for the Primary Endpoint | |
| 5.2.2. Supportive Estimands for the Primary Endpoint | |
| 5.2.3. Estimands for Secondary Endpoints at Week 16 | 17 |
| 5.2.4. Estimands for Secondary Endpoints at Week 24 | 17 |
| 5.3. Adjustments for Covariates | 19 |
| 5.4. Handling of Dropouts or Missing Data | 19 |
| 5.4.1. As Observed Analysis | 20 |
| 5.4.2. Last Observation Carried Forward | 20 |
| 5.4.3. Markov chain Monte Carlo - Multiple Imputation (MCMC- | |
| MI) | |
| 5.5. Multicenter Studies | |
| 5.6. Multiple Comparisons/Multiplicity | |
| 5.7. Patient Disposition. | |
| 5.8. Patient Characteristics | |
| 5.8.1. Demographics and Baseline Characteristics | |
| 5.8.2. Medical History | |
| 5.10. Prior and Concomitant Therapy | |
| 5.11. Efficacy Analyses | |
| 5.12. Health Outcomes/Quality-of-Life Analyses | |
| 5.13. Safety Analyses | 20 |

| J2T-MC-KG | BO (Lebrikizumab) Statistical Analysis Plan Version 2 Pa | ge 3 |
|---|---|---|
| 5.13.1. | Extent of Exposure | 38 |
| 5.13.2. | Adverse Events | 39 |
| 5.13.2.1 | . Common Adverse Events | 40 |
| 5.13.2.2 | Deaths, Other Serious Adverse Events and Other Notable Adverse Events | 40 |
| 5.13.3. | Clinical Laboratory Evaluation | 40 |
| 5.13.4. | Vital Signs and Other Physical Findings | 41 |
| 5.13.5. | Immunogenicity | 41 |
| 5.13.6. | Special Safety Topics including Adverse Events of Special Interest | 43 |
| 5.13.6.1 | . Hepatic Safety | 43 |
| 5.13.6.2 | Eosinophilia and Eosinophil-Related Disorders | 43 |
| 5.13.6.3 | . Infections, including herpes infections and relevant | |
| | parasitic infections | 44 |
| 5.13.6.4 | Conjunctivitis | 44 |
| 5.13.6.5 | . Hypersensitivity | 44 |
| 5.13.6.6 | 5. Injection Site Reactions (ISRs) | 45 |
| 5.13.6.7 | . Malignancies | 45 |
| 5.13.6.8 | Atopic Dermatitis Exacerbation | 45 |
| 5.13.6.9 | 9. Suicide/Self-Injury | 45 |
| 5.14. Subg | group Analyses | 46 |
| 5.15. Proto | ocol Deviations | 46 |
| 5.16. Inter | im Analyses and Data Monitoring | 46 |
| 5.17. Annu | ıal Report Analyses | 47 |
| 5.18. Clini | cal Trial Registry Analyses | 47 |
| 5.19. Biom | narker Analysis | 47 |
| 6. Unblind | ling Plan | 49 |
| 7. Referen | ces | 50 |

## **List of Abbreviations**

| ADA anti-drug antibodies AD atopic dermatitis ADCT Atopic Dermatitis Control Tool AE adverse event AESI adverse events of special interest ALP alkaline phosphatase ALT alanine aminotransferase |
|---|
| ADCT Atopic Dermatitis Control Tool AE adverse event AESI adverse events of special interest ALP alkaline phosphatase |
| AE adverse event AESI adverse events of special interest ALP alkaline phosphatase |
| AESI adverse events of special interest ALP alkaline phosphatase |
| ALP alkaline phosphatase |
| 1 1 |
| ALT alanine aminotransferase |
| AST aspartate transaminase |
| BMI body mass index |
| BSA body surface area |
| CDC Centers for Disease Control and Prevention |
| CDISC Clinical Data Interchange Standards Consortium |
| CDLQI Children's Dermatology Life Quality Index |
| CRF case report form |
| CSR clinical study report |
| CTR Clinical Trial Registry |
| DBL database lock |
| DLQI Dermatology Life Quality Index |
| <b>DSUR</b> Development Safety Update Report |
| EASI Eczema Area and Severity Index |
| <b>EASI-75</b> Eczema Area and Severity Index improvement of ≥75% |
| <b>EASI-90</b> Eczema Area and Severity Index improvement of ≥90% |
| eCRF electronic case report form |
| HLT high-level term |
| ICH International Conference on Harmonisation |

### J2T-MC-KGBO (Lebrikizumab) Statistical Analysis Plan Version 2

Page 6

IGA Investigator's Global Assessment

**ISR** injection site reactions

**Lilly** Eli Lilly and Company

MCMC Markov chain Monte Carlo

MedDRA Medical Dictionary for Regulatory Activities

MI multiple imputation

mTLSS Modified Total Lesion Symptom Scale

**NAb** Neutralizing anti-drug antibodies

NMSC non-melanoma skin cancer

NRS Numeric rating scale

**OI** opportunistic infection

**PD** pharmacodynamic

PhUSE Pharmaceutical Users Software Exchange

**PK** pharmacokinetic

**PROMIS** Patient-Reported Outcomes Information System

PRSQ Participant Reported Satisfaction Question

PT Preferred Term

**Q2W** every 2 weeks

**SAE** serious adverse event

**SAP** statistical analysis plan

**SC** subcutaneously

**SCORAD** SCORing Atopic Dermatitis

**SE** standard error

**SMQ** Standardized MedDRA Query

SOC System Organ Class

TBL total bilirubin

**TE-ADA** treatment-emergent ADA

## J2T-MC-KGBO (Lebrikizumab) Statistical Analysis Plan Version 2

Page 7

**TEAE** treatment-emergent adverse event

**WHO** World Health Organization

WPAI-AD Work Productivity and Activity Impairment Questionnaire-Atopic Dermatitis

# 2. Revision History

Statistical Analysis Plan Version 1 was approved prior to first patient first visit on December 19, 2022.

Changes in Version 2 are documented in the following table. Minor corrections/additions may not be included.

Revisions in SAP Version 2:

| Section | <b>Description of Change</b> | Rationale |
|---|---|---|
| Section 4.1 | Updated the Summary of Study Design to | To account for the Continued Access |
| | reflect KGBO Protocol Addendum 2. | Period. |
| Section 4.3 | Updated to state that participants will | Clarification; this is only a single-arm study |
| | receive Q2W or Q4W dosing after Week | until Week 16. |
| | 16 based on their IGA or EASI score. | |
| Section 5.1.1 | 1. Added Treatment Period II as an | 1. To explicitly define the patient |
| | analysis population to Table 5.1. | population of interest for efficacy analyses after Week 16. |
| | 2. Added text to Table 5.1 to explain | |
| | what analysis populations will be used for each analysis. | 2. Clarification. |
| Section 5.1.2 | Added the baseline period definition for | Clarification. |
| | outcomes collected via eDiary as well as | |
| | what is considered missing. | |
| Section 5.2 | Added a "Primary and Supportive | To clarify the clinical research questions |
| | Estimand" section describing the five | and estimands of interest in this study, and |
| | estimands of interest. | to stay in alignment with LY3650150 |
| | | KGBO(a) Harmonized Clinical Protocol. |
| Section 5.4 | Added how missing data including those | Clarification. |
| | because of intercurrent events will be | |
| | handled for each estimand. | |
| Section 5.4.1. | Removed language explaining how the | This is a single-arm, open-label study until |
| | primary estimand is conditional and not | Week 16 so there is no causal inference no |
| | causal. | matter how the estimand is defined. |
| Section 5.4.2. | 1. Removed the word "sensitivity". | 1. This is a supportive analysis and not a sensitivity analysis. |
| | 2. Added that baseline values will be | |
| | used for imputation if there is no | 2. Clarification. |
| | postbaseline observation. | |
| | | 3. LOCF is only being performed for |
| | 3. Removed the sentence indicating | primary and secondary endpoints. |
| | LOCF will be performed for all | |
| | efficacy data. | |

| Section 5.4.3. | <ol> <li>Removed the term "long-term systemic" from references to rescue medication.</li> <li>Added text to explain that MCMC-MI imputation will be conducted independently for three distinct groups.</li> <li>Added the following 5 endpoints to Table 5.3: Sleep-Loss Scale, Skin Pain NRS, DLQI, cDLQI, and SCORAD.</li> <li>Added a second set of seed numbers to Tabel KGBO.5.3.</li> </ol> | <ol> <li>Rescue medication includes high-potency TCS &gt; 10 days.</li> <li>So that the pattern of missing observations in one treatment group cannot influence missing value imputation in another.</li> <li>MCMC-MI will be performed for all primary and secondary endpoints.</li> <li>MCMC-MI is being performed separately for Weeks 0-16 and Weeks 16-24 of the Treatment Period and therefore requires two different sets of seed numbers.</li> </ol> |
|---|---|---|
| Section 5.8.2. | Updated the eCRF name for both medical history and prespecified medical history. | Correction. |
| Section 5.9 | Updated the names of the eCRF pages that will be used to compute the total number of injections administered. | Correction. |
| Section 5.10 | <ol> <li>Revised the definition of concomitant medication.</li> <li>Added text stating that rescue medications use will be summarized.</li> </ol> | To reflect the addition of the Treatment Period II analysis population. Clarification. |
| Section 5.11 | Added that Pruritus NRS, Skin Pain NRS, and Sleep-Loss Scale will be reported by clinic visit. | Clarification. |
| Section 5.12 | Updated to state that summaries will be provided for the data as-observed and after implementation of LOCF and MCMC-MI imputation. | Data will be presented as-observed and after implementation of LOCF and MCMC-MI imputation for all primary and secondary endpoints. |
| Section 5.13.1 | Updated the name of the eCRF page that will be used to derive the total number of injections received. | Correction. |
| Section 5.13.2 | Added the facial dermatitis follow-up form to Table KGBO.5.5. | Data collected on the facial dermatitis follow-up form will be summarized using descriptive statistics. |
| Section 5.13.3. | Removed scatterplots of baseline-by-<br>maximum values and baseline-by-<br>minimum values from Table KGBO.5.4. | This figure is not required by Version 4 of the Program Safety Analysis Plan. |
| Section 5.13.4. | Removed scatterplots of baseline-by-<br>maximum values and baseline-by-<br>minimum values from Table KGBO.5.4. | This figure is not required by Version 4 of the Program Safety Analysis Plan. |

| Section 5.15 | Updated to state that the primary endpoint, EASI-75, is measured at Week 16. | Clarification. |
|---|---|---|
| Section 5.16 | Added that additional analyses and snapshots of study data may be performed to fulfill the need for regulatory interactions or publication purposes. | To stay in alignment with LY3650150 KGBO(a) Harmonized Clinical Protocol. |
| Appendix 1 | Added definition of rescue medications. | To provide detailed instructions on how to determine rescue medications for this study. |

Abbreviations: AD = atopic dermatitis; CDLQI = Children's Dermatology Life Quality Index; DLQI = Dermatology Life Quality Index; EASI = Eczema Area and Severity Index; LOCF = last observation carried forward; MCMC-MI = Markov chain Monte Carlo-multiple imputation; NRS = numeric rating scale; Q2W = once every 2 weeks; Q4W = once every 4 weeks; SCORAD = SCORing Atopic Dermatitis; TCS = topical corticosteroids.

# 3. Study Objectives

Table KGBO.3.1 shows the protocol-defined objectives and endpoints of the study.

#### Table KGBO.3.1. Protocol-Defined Objectives and Endpoints

#### **Study Primary Objective:**

To evaluate efficacy of lebrikizumab 250 mg Q2W on reducing signs and symptoms of AD at Week 16 in participants with moderate-to-severe AD previously treated with dupilumab

#### **Study Secondary Objective:**

To evaluate the efficacy of lebrikizumab 250 mg Q2W on reducing signs and symptoms of AD at Week 16 and Week 24 in participants with moderate-to-severe AD previously treated with dupilumab

#### **Study Exploratory Objectives**

- To evaluate the efficacy of lebrikizumab 250 mg Q2W in participants with moderate-to-severe AD previously treated with dupilumab
- To discern responder variability within the study and to track response variability to lebrikizumab

#### **Primary Endpoint:**

Percentage of participants achieving EASI-75 at Week 16

#### **Secondary Endpoints:**

- Percentage of participants achieving EASI-75 at Week 24
- Percentage of participants with an IGA score of 0 or 1 and a reduction ≥2 points from baseline to Weeks 16 and 24
- Percentage change in EASI from baseline to Weeks 16 and 24
- Change in EASI from baseline to Weeks 16 and 24
- Percentage of participants achieving EASI-90 from baseline to Weeks 16 and 24
- Percentage of participants with a Pruritus NRS of ≥4 points at baseline who achieve at least 4-point reduction at Weeks 16 and 24
- Percentage of participants with a Pruritus NRS ≥3 points at baseline who achieve at least 3-point reduction at Weeks 16 and 24
- Percentage change in Pruritus NRS score from baseline to Weeks 16 and 24
- Percentage of participants with a Sleep-Loss Scale of ≥2 points at baseline who achieve at least 2-point reduction at Weeks 16 and 24
- Change in Sleep-Loss Scale from baseline at Weeks 16 and 24
- Percentage of participants with a Skin Pain NRS of ≥4 points at baseline who achieve a 4-point reduction from baseline at Weeks 16 and 24
- Change in Skin Pain NRS from baseline to Weeks 16 and 24
- Change in DLQI from baseline to Weeks 16 and Week 24 for participants ≥16 years of age at baseline
- Percentage of participants with at least 4-point at baseline achieving ≥4-point improvement in DLQI from baseline at Weeks 16 and 24 for participants ≥16 years of age at baseline
- Change in cDLQI from baseline to Weeks 16 and 24 for participants <16 years of age at baseline
- Percentage change in SCORAD from baseline to Week 16 and Week 24

#### **Exploratory Endpoints:**

- Percentage change from baseline in mTLss (hands) at Weeks 16 and 24
- Percentage change in ADCT from baseline by visit
- Proportion of TCS/TCI-free days from baseline to Weeks 16 and 24
- Change in body surface area (BSA) from baseline by visit
- Using WPAI-AD by visit, change in baseline in:
  - absenteeism, in those who are currently employed (working for pay)
  - presenteeism, in those who are currently employed (working for pay),

- overall work impairment, in those who are currently employed (working for pay),
- impairment in activities (all participants)
- Percentage of participants with an F-IGA score of 0 or 1 and a reduction ≥2 points from baseline by visit in those who have baseline at least 2 points
- Percentage of participants achieving EASI75 by visit
- Percentage of participants with an IGA score of 0 or 1 and a reduction ≥2 points from baseline by visit
- Percentage change in EASI by visit
- Change in EASI by visit
- Percentage of participants achieving EASI90 by visit
- Percentage of participants with a Pruritus NRS of ≥4 points at baseline who achieve a 4-point reduction by visit
- Percentage of participants with a Pruritus NRS of ≥3 points at baseline who achieve a 3-point reduction by visit
- Percentage change in Pruritus NRS score from baseline by visit
- Percentage of participants with a Sleep-Loss Scale of ≥2 points at baseline who achieve a 2-point reduction by visit
- Change in Sleep-Loss Scale from baseline by visit
- Percentage of participants with a Skin Pain NRS of ≥4 points at baseline who achieve a 4-point reduction from baseline by visit
- Change in Skin Pain NRS from baseline by visit
- Distribution of responses for participant satisfaction (1 question) at Weeks 16 and 24
- Changes from baseline in serum proteins related to AD pathogenesis; Refer to Section 10.2, Appendix 2 of the protocol

# 4. Study Design

### 4.1. Summary of Study Design

Study J2T-MC-KGBO (KGBO) is an open-label, phase 3b study, which is 24 weeks in treatment duration. The study is designed to evaluate the safety and efficacy of lebrikizumab in male and female adult and adolescent participants with moderate-to-severe AD who have been previously treated with dupilumab.

#### **Study Periods**

This trial has 4 study periods:

- Screening (Visit 1: ≤30 days prior to baseline)
- Treatment (Visits 2-9: 24 weeks)
- Safety follow-up (Visit 801: at Week 34 or approximately 12 weeks after last treatment)
- Continued Access (Visits 501, 502, and 503)

Participants who enroll into KGBO Protocol Addendum 2 will move directly into the Continued Access Period after completing the 24-week treatment period. Such participants will not complete Visit 801. A post-treatment follow-up visit (V901) will occur approximately 12 weeks post the last dose at the end of the Continued Access Period for the participants who do not move to commercial lebrikizumab or who discontinued early from the Continued Access Period. Please refer to KGBO Protocol Addendum 2 for more information.

#### **Visit Types**

Study visits at Week 12 (Visit 6) and Week 20 (Visit 8) will be performed virtually, that is, via telephone or telemedicine tools.

All other visits will be conducted at the clinical trial site.

#### **Dosing**

During the 24-week Treatment Period, approximately 120 participants will receive treatment:

- 500 mg subcutaneous (SC) loading dose at baseline and Week 2, followed by 250 mg SC Q2W until Week 16.
- Responders, defined as achieving IGA(0,1) or EASI-75 at Week 16, will receive Q4W dosing and will administer study intervention at Week 20.
- Inadequate responders at Week 16 will receive Q2W dosing and will administer study intervention at Weeks 18, 20, and 22.

During the Continued Access Period, eligible participants will continue lebrikizumab on the same dosing regimen (Q2W or Q4W) they were assigned at Week 16. Please refer to KGBO Protocol Addendum 2 for more information.

The study population is described in Section 5.1.1.

The efficacy and safety assessments are described in Sections 5.11 and 5.13 respectively.

### 4.1.1 Number of Participants

Approximately 120 participants previously treated with dupilumab will be enrolled to study intervention. Among those, approximately 80 participants will be enrolled who discontinued dupilumab due to: a) no response to treatment, b) a partial response to treatment, or c) who lost response to treatment. Additionally, approximately 15 participants will be enrolled who discontinued dupilumab treatment due to intolerance or adverse events (AEs). Finally, approximately 25 participants will be enrolled who stopped dupilumab treatment for other reasons (for example, cost, insurance coverage, access to medication, previous trial participants).

Approximately 10% (n=12) of participants will be adolescents ( $\geq$ 12 to <18 years, weighing  $\geq$ 40 kg). Patients will be evaluated for study eligibility before the baseline visit (Day 1).

#### 4.1.2 Schema

#### Figure KGBO.4.1



Abbreviations: EASI = Eczema Area and Severity Index; IGA = Investigator's Global Assessment; n = number; Q2W = once every 2 weeks; Q4W = once every 4 weeks; SC = subcutaneous; W = week.

<sup>&</sup>lt;sup>a</sup> Weeks 12 and 20 are phone visits.

<sup>&</sup>lt;sup>b</sup> 30-day screening window.

<sup>&</sup>lt;sup>c</sup> Lebrikizumab loading dose of 500 mg SC will be administered at baseline and Week 2.

<sup>&</sup>lt;sup>d</sup> Responders: Participants who reach IGA 0 or 1 (clear or almost clear) or a 75% reduction in the EASI score from baseline (EASI-75). Inadequate responders are participants who do not reach these criteria.

### 4.2. Determination of Sample Size

Based on available data, the anticipated EASI-75 response rate is approximately 50%. A total sample size of 120 enrolled participants will provide >95% probability that the half-width of the 2-sided 90% CI of the EASI-75 response rate is at most 10%.

Example point estimates for EASI-75 response rates and corresponding 2-sided 90% CIs based on the Wilson-Score method for a sample size of 120 participants are summarized in the table below. The CIs are provided as reference rather than a basis of any decision criteria.

Table KGBO.4.1 Estimated 90% CI with Sample Size of 120 Participants

| <b>Example Point Estimates</b> | Lower Bound of 90% CI | Upper Bound of 90% CI |
|---|---|---|
| 40% | 32.9% | 47.5% |
| 45% | 37.7% | 52.5% |
| 50% | 42.6% | 57.4% |
| 55% | 47.5% | 62.3% |
| 60% | 52.5% | 67.1% |

# 4.3. Method of Assignment to Treatment

This is an open-label study. All enrolled patients will be assigned to 250-mg lebrikizumab Q2W at the baseline visit. At Week 16, patients will be assigned to 250-mg lebrikizumab Q2W or 250-mg lebrikizumab Q4W based on their IGA or EASI score.

<sup>&</sup>lt;sup>e</sup> The safety follow-up visit will occur approximately 12 weeks after last study intervention injection.

<sup>&</sup>lt;sup>f</sup> The planned maximum duration of Continued Access treatment will vary for each participant enrolled into KGBO Protocol Addendum 2 and will end if and when the participant meets criteria for discontinuation of study intervention or discontinuation from the study. Participants may remain in the Continued Access Period as long as these criteria for discontinuation are not met and until the sponsor stops the study and addendum.

<sup>&</sup>lt;sup>g</sup> Participants in the Continued Access Period will receive the same dose they were taking during Weeks 16 to 24 of the Treatment Period.

#### 5.A Priori Statistical Methods

#### 5.1. General Considerations

Statistical analysis of this study will be the responsibility of ICON. The latest version of the MedDRA will be used.

Summaries from assessment of endpoints described in the protocol are planned to be included in a CSR. Summaries for key safety data are also planned to be included in the CSR. Results from additional efficacy summaries and other safety summaries may also be provided in the CSR as deemed appropriate.

Any change to the data analysis methods described in the protocol will require a protocol amendment ONLY if it changes a principal feature of the protocol. Any other change to the data analysis methods described in the protocol and the justification for making the change will be described in the CSR.

All statistical processing will be performed using SAS® 9.4 unless otherwise stated.

The schedule of visits and procedures outlined in the protocol specifies the allowable windows for assessments. Assessments performed outside these windows will not be excluded from any summaries, unless specified otherwise.

### 5.1.1. Analysis Populations

Analysis populations are defined in Table KGBO.5.1 along with the analyses they will be used to conduct. The number of patients included in each population will be summarized.

| Table KGBO.5.1. Anal | ysis Popu | lations |
|----------------------|-----------|---------|
|----------------------|-----------|---------|

| Population | Description |
|---|---|
| All Entered Patients | All patients who signed informed consent. Patient flow will be summarized. |
| Intent-to-Treat (ITT) Population | All enrolled patients according to their planned intervention. Unless otherwise specified, efficacy and health outcomes analyses for Weeks 0 to 16 of the Treatment Period will be conducted on this population. |
| Safety Population | All enrolled patients who received at least 1 confirmed dose of lebrikizumab 250 mg. Safety analyses will be conducted on this population. |
| Treatment Period II | All enrolled patients who received at least 1 confirmed dose of lebrikizumab |
| Population | 250 mg during Weeks 16 to 24 of the Treatment Period. Unless otherwise specified, efficacy and health outcomes analyses for Weeks 16 to 24 of the Treatment Period will be conducted on this population. Additional efficacy analyses for Weeks 0 to 24 of the Treatment Period may also be conducted on this population. |

### 5.1.2. General Considerations for Analyses

All analyses will be descriptive. Frequencies, percentages, and 90% Wilson-Score CIs for percentages will be reported for discrete efficacy endpoints. Mean, standard deviation, minimum, Q1, median, Q3, maximum, and the number of participants will be reported for continuous

efficacy endpoints. AEs, discontinuation, and other categorical safety data will be summarized using frequencies and percentages. Continuous vital signs, body weight, and other continuous safety variables including laboratory variables will be summarized descriptively as well.

#### **Baseline**

Baseline will be defined as the last available value before the first injection for efficacy and health outcome analyses. In most cases, this will be the measure recorded at the baseline visit (Day 1). If the patient does not take any injection, the last available value on or prior to treatment assignment date will be used. Change from baseline will be calculated as the visit value of interest minus the baseline value.

For Pruritus Numeric Rating Scale (NRS), Skin Pain NRS, and Sleep-Loss due to Pruritus collected via eDiary, the baseline period is the 7-day window prior to the first injection. A patient must have responses on at least 4 of 7 days to calculate a baseline weekly mean. If a patient has 3 or fewer responses, the baseline mean value will be considered missing.

For the safety analyses, the following baselines will be used. For safety analyses using a baseline period, the baseline period is defined as the time from the screening visit to the date/time of the first injection.

- TEAEs: baseline will be all results recorded during the baseline period.
- Treatment-emergent abnormal laboratory and vital signs results: baseline will be all results recorded during the baseline period.
- Change from baseline to last post-baseline observation or to each scheduled postbaseline visit for laboratory and vital signs results: baseline will be the last scheduled non-missing assessment recorded during the baseline period.

# 5.2. Primary and Supportive Estimands

There will be five estimands addressing different clinical questions of interest and intercurrent events for the primary and secondary endpoints.

### 5.2.1. Primary Estimand for the Primary Endpoint

The primary estimand for the primary endpoint represents the primary clinical question of interest: What is the intervention effect in percentage of participants achieving at least 75% improvement from baseline in Eczema Area and Severity Index (EASI) after 16 weeks of lebrikizumab 250 mg Q2W intervention in participants with moderate-to-severe AD who have been previously treated with dupilumab and who remain on study treatment until Week 16?

The primary estimand for the primary endpoint is described by the following attributes:

- A. Population: participants with moderate-to-severe AD who have been previously treated with dupilumab and who remain on study treatment until Week 16.
- B. Endpoint: whether participants achieve at least 75% improvement from baseline in EASI at Week 16.

- C. Intercurrent events: There are no intercurrent events for this population since participants who initiate rescue medication are discontinued from the study and hence study treatment. Therefore, participants who stay on study treatment through Week 16 will not have an intercurrent event such as initiating rescue medication or permanently discontinuing treatment.
- D. Population-level summary: percentage of participants achieving EASI-75 response at Week 16.

### 5.2.2. Supportive Estimands for the Primary Endpoint

There are two supportive estimands for the primary endpoint. The first is a hybrid estimand representing the following clinical question of interest: What is the intervention effect in percentage of participants achieving at least 75% improvement from baseline in Eczema Area and Severity Index (EASI) after 16 weeks of lebrikizumab 250 mg Q2W intervention in participants with moderate-to-severe AD who have been previously treated with dupilumab if all participants adhered to treatment except those who discontinued due to lack of efficacy?

This estimand is described by the following attributes:

- A. Population: participants with moderate-to-severe AD who have been previously treated with dupilumab.
- B. Endpoint: whether participants achieve at least 75% improvement from baseline in EASI at Week 16.
- C. Intercurrent events (ICEs): One ICE, permanent treatment discontinuation, is considered by this estimand as follows:
  - a. Participants who discontinue treatment due to lack of efficacy prior to Week 16 will be considered as treatment failures, i.e. non-responders, after the ICE. Therefore, a composite strategy is used for this type of ICE.
  - b. For participants who discontinue treatment due to reasons other than lack of efficacy prior to Week 16, a hypothetical strategy will be used to estimate what the treatment effect would have been if subjects continued with treatment. Therefore, a hypothetical strategy is used for this type of ICE.
- D. Population-level summary: percentage of participants achieving EASI-75 response at Week 16.

The second supportive estimand for the primary endpoint is a hypothetical estimand representing the following clinical question of interest: What is the intervention effect in percentage of participants achieving at least 75% improvement from baseline in Eczema Area and Severity Index (EASI) after 16 weeks of lebrikizumab 250 mg Q2W intervention in participants with moderate-to-severe AD who have been previously treated with dupilumab if all participants adhered to treatment?

This estimand is described by the following attributes:

A. Population: participants with moderate-to-severe AD who have been previously treated with dupilumab.

- B. Endpoint: whether participants achieve at least 75% improvement from baseline in EASI at Week 16.
- C. Intercurrent events (ICEs): One ICE, permanent treatment discontinuation, is considered by this estimand as follows:
  - a. For participants who discontinue treatment prior to Week 16, a hypothetical strategy will be used to estimate what the treatment effect would have been if all subjects continued with treatment. Therefore, a hypothetical strategy is used for this type of ICE.
- D. Population-level summary: percentage of participants achieving EASI-75 response at Week 16.

### 5.2.3. Estimands for Secondary Endpoints at Week 16

The primary estimand for the primary endpoint will be applied to all secondary endpoints at Week 16. The supportive estimands for the primary endpoint will also be applied to all secondary endpoints at Week 16.

### 5.2.4. Estimands for Secondary Endpoints at Week 24

The primary estimand for the primary endpoint will be applied to all secondary endpoints at Week 24. There are two supportive estimands for secondary endpoints at Week 24. The first is a hybrid estimand representing the following clinical question of interest: What is the intervention effect in successful responses or means after 24 weeks of lebrikizumab intervention in participants with moderate-to-severe AD who have been previously treated with dupilumab if all participants adhered to treatment except those who discontinued due to lack of efficacy?

This estimand is described by the following attributes:

- A. Population: Treatment Period II population as described in Section 5.1.1.
- B. Endpoint: apply to all secondary endpoints at Week 24.
- C. Intercurrent events (ICEs): One ICE, permanent treatment discontinuation, is considered by this estimand as follows:
  - a. Participants who discontinue treatment due to lack of efficacy after Week 16 will be considered as treatment failures, i.e. non-responders, after the ICE. Therefore, a composite strategy is used for this type of ICE.
  - b. For participants who discontinue treatment due to reasons other than lack of efficacy after Week 16, a hypothetical strategy will be used to estimate what the treatment effect would have been if subjects continued with treatment. Therefore, a hypothetical strategy is used for this type of ICE.
- D. Population-level summary: percentage of successful responses or means at Week 24.

The second supportive estimand for secondary endpoints at Week 24 is a hypothetical estimand representing the following clinical question of interest: What is the intervention effect in successful responses or means after 24 weeks of lebrikizumab 250 mg Q2W intervention in

participants with moderate-to-severe AD who have been previously treated with dupilumab if all participants adhered to treatment?

This estimand is described by the following attributes:

- A. Population: Treatment Period II population as described in Section 5.1.1.
- B. Endpoint: apply to all secondary endpoints at Week 24.
- C. Intercurrent events (ICEs): One ICE, permanent treatment discontinuation, is considered by this estimand as follows:
  - a. For participants who discontinue treatment after Week 16, a hypothetical strategy will be used to estimate what the treatment effect would have been if all subjects continued with treatment. Therefore, a hypothetical strategy is used for this type of ICE.
- D. Population-level summary: Population-level summary: percentage of successful responses or means at Week 24.

Because participants who initiate rescue medication are required to discontinue from the study and hence permanently discontinue study treatment, the supportive estimands for the primary and secondary endpoints only consider permanent treatment discontinuation as an ICE.

Analytical details on how missing data including those as a result of intercurrent events will be handled can be found in Section 5.4. The following table (Table KGBO.5.2) summarizes the analytical strategies that will be conducted on the intercurrent events for the five estimands.

**Table KGBO.5.2. Description of Primary and Supportive Estimands** 

| | | Analysis Strategy for the ICE of<br>Permanent Treatment<br>Discontinuation | | Missing<br>Data |
|---|---|---|---|---|
| Estimand | Population | Due to lack of efficacy | Due to any other<br>reasons, including<br>initiation of rescue<br>medication | Imputation<br>Method |
| Primary Estimand<br>for the Primary<br>Endpoint and<br>Secondary<br>Endpoints | ITT Population<br>who remained on<br>treatment | Not applicable | Not applicable | Primary<br>analysis: as<br>observed |
| Supportive Estimand for the Primary Endpoint and Secondary | ITT Population | Composite:<br>Set to baseline | Hypothetical: Set to missing | MCMC-MI |

| Endpoints at Week<br>16 (Hybrid) | | | | |
|---|---|---|---|---|
| Supportive Estimand for the Primary Endpoint and Secondary Endpoints at Week 16 (Hypothetical) | ITT Population | Hypothetical:<br>Set to missing | Hypothetical: Set to missing | LOCF |
| Supportive Estimand for Secondary Endpoints at Week 24 (Hybrid) | Treatment Period II Population | Composite:<br>Set to baseline | Hypothetical: Set to missing | MCMC-MI |
| Supportive Estimand for Secondary Endpoints at Week 24 (Hypothetical) | Treatment Period II Population | Hypothetical:<br>Set to missing | Hypothetical: Set to missing | LOCF |

Abbreviations: ICE = intercurrent event; LOCF = last observation carried forward; MCMC = Markov chain Monte Carlo; MI = Multiple Imputation.

### 5.3. Adjustments for Covariates

No statistical tests will be performed.

# 5.4. Handling of Dropouts or Missing Data

Intercurrent events, as per the ICH guideline (ICH E9R1), are events which occur after the treatment initiation and make it impossible to measure a variable or influence how it should be interpreted. Examples of such events include treatment discontinuation due to death or AEs, rescue treatment, and loss to follow-up.

This section describes missing data imputation methods handling intercurrent events, which will be implemented in this study. For efficacy analyses relative to the primary estimand for primary and secondary endpoints, the method of handling missing data will be the "as observed" strategy described in Section 5.4.1.

For efficacy analyses relative to the supportive hypothetical estimands for primary and secondary endpoints, missing data including those because of intercurrent events will be imputed using the Last Observation Carried Forward (LOCF) strategy described in Section 5.4.2.

For efficacy analyses relative to the supportive hybrid estimands for primary and secondary endpoints, missing data including those because of intercurrent events will be imputed using Markov Chain Monte Carlo Multiple Imputation (MCMC-MI) as described in Section 5.4.3.

### 5.4.1. As Observed Analysis

The "as observed" strategy is used in so-called "observed cases" or "completers" analysis ubiquitous in the literature. For this analysis, only data from completers at the visit are relevant. All efficacy data will be summarized using an "as observed" analysis and summaries based on observed data at each postbaseline visit will be provided.

#### 5.4.2. Last Observation Carried Forward

In this analysis, all missing values will be imputed using last observation carried forward (LOCF). Baseline values will be used for imputation if there is no postbaseline observation.

### 5.4.3. Markov Chain Monte Carlo - Multiple Imputation (MCMC-MI)

The method of handling missing efficacy data relative to the supportive hybrid estimands for the primary and secondary endpoints at Week 16 will be based on Markov Chain Monte Carlo Multiple Imputation (MCMC-MI). For patients who discontinue treatment due to lack of efficacy prior to Week 16, set to the patient's baseline value subsequent to this time through Week 16. MCMC-MI will be used to handle the remaining missing data.

The method of handling missing efficacy data relative to the supportive hybrid estimand for secondary endpoints at Week 24 will be based on MCMC-MI. For patients who discontinue treatment due to lack of efficacy after Week 16, set to the patient's baseline value subsequent to this time through Week 24. MCMC-MI will be used to handle the remaining missing data. Imputation will be conducted within each treatment group independently so that the pattern of missing observations in one treatment group cannot influence missing value imputation in another.

For each imputation process, 25 datasets with imputations will be calculated. The initial seed values are given in Table KGBO.5.3. The response rates and their associated SEs will be computed for each data set using SAS PROC FREQ with the riskdiff option specified for the appropriate column in the TABLES statement. The response rates and SEs from the resulting output will be combined across the 25 imputed datasets using SAS PROC MIANALYZE.

For binary responses related to EASI and IGA, the binary response variables will be calculated based on the multiply imputed datasets that have been created. Because the MCMC algorithm is based on the multivariate normal model, imputed values for IGA will not generally be one of the discrete values used in IGA scoring (0, 1, 2, 3, or 4). Therefore, to derive the binary IGA response variable, standard rounding rules will be applied to the imputed values. For example, if a patient has an IGA score imputed as 1.4 (and assuming a baseline IGA score of 3), the imputed value would be rounded down to 1, and the minimum change from baseline of 2 would have been met. This patient would be considered a responder.

For derivation of an EASI-75 and EASI-90 response, no rounding will be performed. The imputed EASI value will be compared directly to the observed baseline EASI value to determine whether a reduction of at least 75% or 90% was achieved at each visit.

For derivation of the following Pruritus NRS, Skin Pain NRS, Sleep-Loss Scale, and DLQI responses, no rounding will be performed. The imputed Pruritus NRS, Skin Pain NRS, and Sleep-Loss Scale values will be compared directly to the observed mean baseline values to determine whether a response was achieved. The imputed DLQI values will be compared directly to the observed baseline values to determine whether a response was achieved.

- Proportion of patients with a Pruritus NRS of ≥3 points at baseline achieving at least a 3-point reduction by visit.
- Proportion of patients with a Pruritus NRS of ≥4 points at baseline achieving at least a 4-point reduction by visit.
- Proportion of patients with a Skin Pain NRS of ≥4 points at baseline achieving at least a 4-point reduction by visit.
- Proportion of patients with a Sleep-Loss Scale of ≥2 points at baseline achieving at least a 2-point reduction by visit.
- Proportion of patients with DLQI of ≥4 points at baseline achieving at least a 4-point reduction by visit.

Note that the estimate and 90% confidence interval bounds output by this SAS PROC MIANALYZE are percents (i.e, they are in terms of the response rate). To obtain the number of responders, the estimated percent is multiplied by the number of individuals in the analysis population and rounded to the nearest integer.

Imputation of continuous data will parallel that of binary variables. IGA, EASI, Sleep-Loss, Skin Pain NRS, Pruritus NRS, DLQI, CDLQI, and SCORAD will be summarized using an MCMC-MI analysis.

**Table KGBO.5.3. Seed Values for MCMC-Multiple Imputation** 

| Analysis | Seed Values for Weeks 0-<br>16 of the Treatment<br>Period;<br>LEB 250mg Q2W | Seed Values for Weeks 16-<br>24 of the Treatment Period;<br>LEB 250mg Q2W or Q4W |
|---|---|---|
| Proportion of patients achieving IGA of 0 or 1 with a $\geq 2$ -point improvement from baseline by visit. | 661769200 | 893745627 |
| Percent change from baseline in EASI score by visit. EASI-75 and EASI-90 will leverage imputation from EASI and therefore use the same seed numbers. | 153233047 | 345987238 |
| Change from baseline in Pruritis NRS Score by visit. Proportion of patients with a Pruritus NRS Score of ≥3 or ≥4 points at baseline achieving at least a 3point or 4-point reduction will leverage imputation from Pruritis NRS Score and therefore use the same seed numbers. | 502899349 | 302781834 |
| Change from baseline in Sleep-Loss Scale by visit. Proportion of patients with a Sleep-Loss Scale of ≥2 points at baseline who achieve at least a 2-point reduction at each visit will leverage imputation from Sleep-Loss Scale and therefore use the same seed numbers. | 691405299 | 999692612 |
| Change from baseline in Skin Pain NRS from baseline by visit. Proportion of patients with a Pruritus NRS Score of ≥4 points at baseline achieving at least a 4-point reduction will leverage imputation from Pruritis NRS Score and therefore use the same seed numbers. | 81969225 | 20532740 |
| Change from baseline in DLQI by visit. Proportion of patients with DLQI ≥4 points at baseline achieving at least a 4-point reduction will leverage imputation from DLQI and therefore use the same seed numbers. | 66350097 | 60458639 |
| Change from baseline in CDLQI by visit. | 93794487 | 34792746 |
| Change from baseline in SCORAD by visit. | 90372454 | 71154457 |

Abbreviations: CDLQI = Children's Dermatology Life Quality Index; DLQI = Dermatology Life Quality Index; EASI = Eczema Area and Severity Index; EASI-75 = Eczema Area and Severity Index improvement of ≥75%; EASI-90 = Eczema Area and Severity Index improvement of ≥90%; IGA = Investigator's Global Assessment for Atopic Dermatitis; LEB = lebrikizumab; MCMC = Markov chain Monte Carlo; NRS = Numeric Rating Scale; Q2W = every 2 weeks; Q4W = every 4 weeks; SCORAD = SCORing Atopic Dermatitis.

#### 5.5. Multicenter Studies

This study will be conducted by multiple investigators at multiple sites.

### **5.6. Multiple Comparisons/Multiplicity**

No statistical tests will be performed in this study so there is no need to account for multiple comparisons.

### 5.7. Patient Disposition

The following patient disposition summaries will be provided (details of the analysis populations can be found in Section 5.1.1):

- The total number and percentage of patients entering each statistical analysis population as defined in Section 5.1.1 (analysis population: all entered patients).
- The number and percentage of patients who entered the study, were treated, and screen failed will be provided overall and by screen fail reason (analysis population: all entered patients).
- The number and percentage of patients who completed Week 16, and the number and percentage of patients who discontinued the treatment at any time before Week 16, by primary reason for discontinuation of treatment (analysis population: ITT).
- The number and percentage of patients who completed Week 24, and the number and percentage of patients who discontinued the treatment at any time before Week 24, by primary reason for discontinuation of treatment (analysis population: ITT).
- The number and percentage of patients who were treated and completed the study, and the number and percentage of patients who discontinued the study at any time, by primary reason for discontinuation (analysis population: ITT).

All enrolled participants (that is, in the ITT population) who discontinued from study treatment will be listed together with the discontinuation reason, and the timing of discontinuation from the study will be reported.

Patient allocation by center/site will be summarized with the number of patients who entered the study, number of ITT patients, number of patients discontinued from study treatment, and number of patients discontinued from the study.

#### 5.8. Patient Characteristics

# 5.8.1. Demographics and Baseline Characteristics

Patient demographic variables and baseline characteristics will be summarized for the ITT and Treatment Period II populations. The continuous variables will be summarized using descriptive statistics (mean, median, standard deviation, and range [minimum and maximum]), and the categorical variables will be summarized using frequency counts and percentages.

The following demographic information will be included:

- age
- sex (male, female)
- reason of prior dupilumab discontinued
- Fitzpatrick skin phototype
- race (American Indian or Alaska Native, Asian, Black or African American, Native Hawaiian or Other Pacific Islander, White, Multiple, Other, or Not Reported)
- ethnicity (Hispanic or Latino, Not Hispanic or Latino, Not reported, or Unknown)
- weight (kg)
- weight category  $(40-<60 \text{ kg}, \ge 60 \text{ to } <100 \text{ kg}, \text{ or } \ge 100 \text{ kg})$
- height (cm)
- BMI (kg/m<sup>2</sup>), and
- BMI category (Underweight [ $<18.5 \text{ kg/m}^2$ ], Normal [ $\ge18.5 \text{ and } <25 \text{ kg/m}^2$ ], Overweight [ $\ge25 \text{ and } <30 \text{ kg/m}^2$ ], Obese [ $\ge30 \text{ and } <40 \text{ kg/m}^2$ ], or Extreme obese [ $\ge40 \text{ kg/m}^2$ ]).

By-patient listings of basic demographic information for the ITT population will be provided.

The following baseline disease/clinical characteristics will be included:

- age at onset (years): calculated as the difference between date of onset of AD and the date of birth collected on the CRF
- duration since AD onset (years): calculated as the difference between date of informed consent and the date of onset of AD collected on the CRF
- duration since AD onset category (0 to <2 years, 2 to <5 years, 5 to <10 years, or ≥10 years)
- anatomical area affected by AD:
  - head
  - o trunk (internal/medial axillae and groin)
  - o upper extremities (includes external axillae)
  - o lower extremities (includes buttocks and feet), and
  - o at least 2 areas
- AD treatment used in the past:
  - o none
  - o topical corticosteroids
  - o topical calcineurin inhibitors

o immunosuppressive/immunomodulating drugs: systemic corticosteroids, cyclosporine, mycophenolate-mofetil, IFN-γ, janus kinase inhibitors, azathioprine, methotrexate, phototherapy, photochemotherapy, and other biologics (eg, B-cell depleting biologics)

The following efficacy instruments will be included:

- IGA
- F-IGA score
- EASI score
- BSA
- SCORAD
- mTLSS
- Pruritus NRS
- Sleep-Loss Scale
- Skin Pain NRS
- DLQI/CDLQI
- ADCT
- Participant-Reported Satisfaction Question
- Fitzpatrick Skin Phototype Assessment
- WPAI-AD.

# 5.8.2. Medical History

Medical histories are defined as the conditions/events recorded on the *Pre-existing Conditions* and *Medical History* eCRF with a start date prior to the first study drug injection. Notice if a medical history worsens in severity on or after the date of first injection it will be recorded as an AE on the *Adverse Event* eCRF with the date of worsening as the start date.

The number and percentage of patients with medical histories will be summarized for the ITT population using the MedDRA Preferred Term (PT) nested within System Organ Class (SOC).

The number and percentage of patients with specific medical history events of interest prespecified on the *Prespecified Medical History* eCRF will be summarized for the ITT population.

# 5.9. Treatment Compliance

Beginning Week 4 (Visit 4) the participant/caregiver will be encouraged to administer the study intervention while in the clinic or at home. Participants may choose to continue to receive study drug injections administered by trained clinic staff for any visit occurring in the clinic. Home

dosing must be self-administered or given by a caregiver that has received proper injection technique training.

When participants self-administer study intervention(s) at home, compliance with study intervention will be assessed at each visit. Compliance will be assessed by direct questioning, counting returned injection supplies, and documented in the source documents.

Treatment compliance with investigational product will be summarized for patients who receive at least 1 confirmed dose of lebrikizumab (ie, the Safety Population) during the Treatment Period. Treatment compliance for each patient will be calculated as:

Treatment compliance (%) = 
$$100 \times \frac{Total\ number\ of\ injections\ administered}{Total\ number\ of\ injections\ expected}$$

- The number of injections expected can be derived from the study drug dispense dataset.
- The total number of injections administered will be based on the *Exposure as Collected* eCRF page and on the *Exposure as Collected: Missed Injections at Home* eCRF page.

A patient will be considered compliant if he or she received ≥75% of the expected number of injections while enrolled in the study. Descriptive statistics for percent compliance will be summarized. Subintervals of interest, such as compliance between visits, may also be presented.

### 5.10. Prior and Concomitant Therapy

Medications will be classified into anatomical therapeutic chemical (ATC) drug classes using the latest version of the World Health Organization (WHO) drug dictionary. Medication start and stop dates will be compared to the date of first dose of treatment during Weeks 0-16 of the Treatment Period and Weeks 16-24 of the Treatment Period to be classified as concomitant for each treatment period.

Prior medications are those medications that start and stop prior to the date of first dose of study treatment. Concomitant medications are those medications that start before, on, or after the first day of study treatment of the defined study period (that is, Weeks 0-16 or Weeks 16-24 of the Treatment Period) and continue into that period. Concomitant medications are assigned to the study period in which they are actually ongoing. For example, if a participant is receiving a concomitant medication during Weeks 0-16 but has a stop date prior to Week 16, the same medication would not be listed as a concomitant medication for Weeks 16-24 unless the patient has a new start date.

Prior medication will be summarized by drug class and PT for the ITT population. Concomitant medication used during Weeks 0-16 and Weeks 16-24 will be presented separately for the ITT and Treatment Period II populations.

Rescue medications used during Weeks 0-16 and Weeks 16-24 will be presented separately for the ITT and Treatment Period II populations. This will include: (1) topical therapy and (2) systemic therapy (e.g., systemic corticosteroids, phototherapy, cyclosporin, etc.). More information on the definition of rescue medications can be found in Appendix 1.

# 5.11. Efficacy Analyses

<u>Table KGBO.5.4</u> includes the description and derivation of the efficacy measures and endpoints.

For categorical parameters, the number and percentage of patients in each category will be presented, as well as a 90% Wilson-Score confidence interval for the percentage. For continuous parameters, descriptive statistics will include n (number of patients), mean, standard deviation, Q1, median, Q3, minimum, and maximum. These summaries will be provided for the data as-observed and after implementation of LOCF and MCMC-MI imputation as described in Sections 5.4.2 and 5.4.3.

The IGA, F-IGA, EASI, BSA, Pruritus NRS, Skin Pain NRS, and Sleep-Loss Scale will be reported by clinic visit.

### Table KGBO.5.4.Description and Derivation of Efficacy/Health Outcomes Measures and Endpoints

| | | | | T |
|---|---|---|---|---|
| Measure | Description | Variable | Derivation/Comment | Imputation Approach if<br>Missing Components |
| Investigator's | The IGA is a static assessment and rates | IGA score | Single item. Range: 0-4 | Single item, missing if |
| Global | the severity of a patient's AD. The IGA | | 0 represents "clear" | missing |
| Assessment | is comprised of a 5-point scale ranging | | 4 represents "severe" | |
| (IGA) | from 0 (clear) to 4 (severe), and a score | • IGA (0,1) with | Observed score of 0 or 1 and | Missing if baseline or |
| | is selected using descriptors that best describe the overall appearance of the | ≥2-point improvement <sup>a</sup> | change from baseline ≤-2 | observed value is missing |
| | lesions at a given time point. | IGA (0) | Observed score of 0 | Single item, missing if missing |
| Face- | The F-IGA is a static assessment and | F-IGA Score | Single item. Range: 0-4, 0 represents | Single item, missing if |
| Investigator's | rates the severity of a patient's AD on | | "clear", 4 represents "severe" | missing |
| Global | the face. The F-IGA is comprised of a | IGA $(0,1)$ with $\geq 2$ -point | Observed score of 0 or 1 and change | Missing if baseline or |
| Assessment (F-IGA) | 5-point scale ranging from 0 (clear) to 4 (severe), and a score is selected using | improvement <sup>a</sup> | from baseline ≤-2 | observed value is missing |
| | descriptors that best describe the overall | IGA (0) | Observed score of 0 | Single item, missing if |
| | appearance of the lesions at a given time point. | | | missing |
| Eczema Area | The EASI scoring system uses a defined | EASI score | Derive EASI region score for each of | NA: partial assessments |
| and Severity | process (Steps 1-5 below) to grade the | | head and neck, trunk, upper limbs, and | cannot be saved. |
| Index | severity of the signs of eczema and the | | lower limbs as follows: | |
| (EASI) | extent affected. The extent of disease | | EASI <sub>region</sub> = (erythema + | |
| | (percentage of skin affected: $0 = 0\%$ ; | | edema/papulation + excoriation + | |
| | 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; | | lichenification)*(value from percentage | |
| | 4 = 50-69%; 5 = 70-89%; 6 = 90-100%) | | involvement), where erythema, | |
| | and the severity of 4 clinical signs | | edema/papulation, excoriation, and | |
| | (erythema, edema/papulation, | | lichenification are evaluated on a scale | |
| | excoriation, and lichenification) each on | | of 0 to 3, and value from percentage | |
| | a scale of 0-3 ( $0 = \text{none}$ , absent; | | involvement is on a scale of 0 to 6. | |
| | $1 = \text{mild}$ ; $2 = \text{moderate}$ ; $3 = \text{severe}$ ) at $\underline{4}$ | | Then total EASI score is as follows: | |

| | body sites (head and neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. Each body site will have a score that ranges from 0-72, and the final EASI score will be obtained by weight-averaging these 4 scores. Hence, the final EASI score will range from 0-72 for each time point. | Change from baseline in EASI score Percent change from baseline EASI score <sup>a</sup> | $EASI = 0.1*EASI_{head \ and \ neck} + \\ 0.3*EASI_{trunk} + 0.2*EASI_{upper \ limbs} + \\ 0.4*EASI_{lower \ limbs}$ Change from baseline: observed EASI score $Change from \ baseline: absolute the score of the second of the sec$ | Missing if baseline or observed value is missing |
|---|---|---|---|---|
| | | EASI-75a | % improvement in EASI score from baseline ≥75%: % change from baseline ≤-75 | Missing if baseline or observed value is missing |
| | | EASI-90a | % improvement in EASI score from baseline ≥90%: % change from baseline ≤-90 | Missing if baseline or observed value is missing |
| Body Surface<br>Area (BSA)<br>Affected by | The BSA assessment estimates the extent of disease or skin involvement with respect to AD and is expressed as a | BSA score | $\begin{aligned} BSA \ Total &= BSA_{head \ and \ neck} + \\ BSA_{trunk} + BSA_{upper \ limbs} + BSA_{lower} \\ \\ limbs \end{aligned}$ | NA: partial assessments cannot be saved. |
| AD | percentage of total body surface. BSA will be determined by the investigator or designee using the patient palm = 1% rule. | Change from baseline in BSA score <sup>a</sup> | Change from baseline: observed BSA score - baseline BSA score | Missing if baseline or observed value is missing. |
| Dermatology<br>Life Quality<br>Index (DLQI) | The DLQI is a validated, dermatology-specific, patient-reported measure that evaluates a patient's HRQoL. This questionnaire has 10 items that are grouped in 6 domains, including symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. The recall | DLQI total score | A DLQI total score is calculated by summing all 10 question responses and has a range of 0-30 (less to more impairment) (Finlay and Khan 1994; Basra et al. 2008). | Score of 1 unanswered question = 0; If 2 or more questions are missing, the total score is missing. Note: #7B could be a valid missing while #7A is not "No." That is, #7 should be considered as 1 question. |
| | period of this scale is over the "last week". | DLQI (0,1) | A DLQI (0,1) response is defined as a postbaseline DLQI total score of 0 or 1. A DLQI total score of 0-1 is considered as having no effect on a patient's | Missing if DLQI total score is missing |

| Response categories and corresponding scores are: | | HRQoL (Khilji et al. 2002; Hongbo et al. 2005). | |
|---|---|---|---|
| Very much = 3<br>A lot = 2 | 4-point improvementa | Change from baseline ≤-4 | Missing if baseline is missing or observed value is |
| A lot $\frac{1}{2}$ | | | missing. |
| Not at all = 0 | DLQI total score and | Calculated as: observed DLQI (total | Missing if baseline or |
| Not relevant = 0 | domain scores change<br>from baseline <sup>a</sup> | score or domain scores) - baseline DLQI (total score or domain scores) | observed value is missing |
| Scores range from 0-30, with higher | | , | |
| scores indicating greater impairment of | | | |
| QoL. A DLQI total score of 0-1 is | | | |
| considered as having no effect on a | | | |
| patient's HRQoL (Hongbo et al. 2005), | | | |
| and a 4-point change from baseline is | | | |
| considered as the minimal clinically | | | |
| important difference threshold (Khilji et | | | |
| al. 2002; Basra et al. 2015). | | | |
| | DLQI symptoms and | Sum of responses of questions 1 and 2: | If 1 question in a domain is |
| | feelings domain | 1. How itchy, sore, painful or stinging | missing, that domain is |
| | | has your skin been? | missing. |
| | | 2. How embarrassed or self-conscious | |
| | | have you been because of your | |
| | DI OL 1. 'lea esties't' | skin? | IC1 |
| | DLQI daily activities domain | Sum of responses of questions 3 and 4: | If 1 question in a domain is |
| | domain | 3. How much has your skin interfered with you going shopping or looking | missing, that domain is missing. |
| | | after your home or garden? | missing. |
| | | 4. How much has your skin influenced | |
| | | the clothes you wear? | |
| | DLQI leisure domain | Sum of responses of questions 5 and 6: | If 1 question in a domain is |
| | | 5. How much has your skin affected any | missing, that domain is |

| | | DLQI work and school domain | social or leisure activities? 6. How much has your skin make it difficult for you to do any sport? Sum of responses of questions 7A and 7B: 7A. Has your skin prevented you from working or studying? | If the answer to question 7A is missing, this domain is missing. If 7A is No, and 7B is missing, this domain |
|---|---|---|---|---|
| | | | 7B. If No: how much has your skin been a problem at work or studying? | is missing. |
| | | DLQI personal relationships domain | Sum of responses of questions 8 and 9: 8. How much has your skin created problems with your partner or any of your close friends or relatives? 9. How much has your skin caused any sexual difficulties? | If 1 question in a domain is missing, that domain is missing. |
| | | DLQI treatment domain | Response of question 10: 10. How much of a problem has the treatment for your skin been, for example by making your home messy, or by taking up time? | If 1 question in a domain is missing, that domain is missing. |
| Dermatology Life Quality Index (CDLQI) The scon Very Quit Only Not | The CDLQI is designed to measure the impact of any skin disease on the lives of children. Patients ≤16 years will complete the CDLQI and should continue to complete the CDLQI for the duration of the study. The scoring of each question is: | CDLQI total score | A CDLQI total score is calculated by summing all 10 question responses and has a range of 0-30 (less to more impairment) (Waters A et al. 2010). | Score of 1 unanswered<br>question = 0; If 2 or more<br>questions are missing, the<br>total score is missing. |
| | | CDLQI (0,1) | A CDLQI (0,1) response is defined as a postbaseline CDLQI total score of 0 or 1. | Missing if CLQI total score is missing |
| | • Very much = 3 | 4-point improvement <sup>a</sup> | Change from baseline ≤-4 | Missing if baseline or observed value is missing |
| | <ul><li>Only a little = 1</li><li>Not at all = 0</li></ul> | CDLQI total score and<br>domain scores change<br>from baseline <sup>a</sup> | Calculated as: observed CDLQI (total score or domain scores) - baseline CDLQI (total score or domain scores) | Missing if baseline or observed value is missing |
| | | CDLQI symptoms and feelings domain | Sum of responses of questions 1 and 2: 1. Over the last week, how itchy, | If 1 question in a domain is missing, that domain is |

| • Question 7: 'Prevented school' (text-only questionnaire) = 3 | | "scratchy", sore or painful has your skin been? 2. Over the last week, how embarrassed or self conscious, upset or sad have you been because of your skin? | missing. |
|---|---|---|---|
| | CDLQI sleep domain | Response of question 9 9. Over the last week, how much has your <b>sleep</b> been affected by your skin problem? | Single item, missing if missing |
| | CDLQI leisure domain | 6: 4. Over the last week, how much have you changed or worn different or special clothes/shoes because of your skin? 5. Over the last week, how much has your skin trouble affected going out, playing, or doing hobbies? 6. Over the last week, how much have you avoided swimming or other sports because of your skin trouble? | If 1 question in a domain is missing, that domain is missing. |
| | CDLQI school or<br>holiday domain | Responses of questions 7: If select 'Prevented school', score = 3 | Single item, missing if missing |
| | | | Last week. was it school time? OR was it holiday time? | If school time: Over the last week, how much did your skin affect your school work? If holiday time: How much over the last week, has your skin problem interfered with your enjoyment of the holiday? | |
|---|---|---|---|---|---|
| | | CDLQI personal relationships domain | you names, teas | c, how much has ed your c, how much had because of ther people calling | If 1 question in a domain is missing, that domain is missing. |
| | | CDLQI treatment domain | Response of question<br>10. How much of a partent treatment for you | problem has the | Single item, missing if missing. |
| SCORing<br>Atopic<br>Dermatitis<br>(SCORAD) | SCORAD is a validated clinical tool for assessing the extent and intensity of atopic dermatitis. There are 3 components to the assessment: • The extent of AD is assessed as a percentage of each | SCORAD Score | SCORAD = $A/5 + 7$<br>A is extent of disease<br>B is disease severity<br>C is subjective symp | e, range 0-100<br>, range 0-18 | Missing if components A and B are missing or if component C is missing. Partial assessments performed by physician cannot be saved and partial |

| | defined body area and<br>reported as the sum of all<br>areas, with a maximum score | Change from baseline | Change from baseline: observed | assessments performed by subject cannot be saved. |
|---|---|---|---|---|
| | of 100% (assigned as "A" in<br>the overall SCORAD<br>calculation). | in SCORAD score | SCORAD score – baseline SCORAD score | Missing if baseline or observed value is missing. |
| | The severity of 6 specific symptoms of AD (redness, swelling, oozing/crusting, excoriation, skin | Percent change from<br>baseline in SCORAD<br>score | % change from baseline: $100 \times \frac{Observed\ score - Baseline}{Baseline}$ | |
| | thickening/lichenification,<br>dryness) is assessed using the<br>following scale: none (0),<br>mild (1), moderate (2), or | SCORAD75 | % Improvement in SCORAD from baseline ≥75%: % change from baseline ≤-75 | Missing if baseline or observed value is missing. |
| | severe (3) (for a maximum of 18 total points, assigned as "B" in the overall SCORAD calculation). | SCORAD90 | % Improvement in SCORAD from baseline ≥90%: % change from baseline ≤-90 | Missing if baseline or observed value is missing. |
| | <ul> <li>Subjective assessment of itch<br/>and of sleeplessness is<br/>recorded for each symptom by<br/>the patient or relative on a</li> </ul> | | | |
| | VAS, where 0 is no itch (or sleeplessness) and 10 is the | | | |
| | worst imaginable itch (or sleeplessness), with a maximum possible score of 20 | | | |
| | (assigned as "C" in the overall SCORAD calculation. | | | |
| Modified | The Modified Total Lesion Symptom | Percent change from | This composite score assigns 0 (mild) to | If 1 question in a domain is |
| Total Lesion Symptom | Scale is an investigator-reported scale that combines the evaluation of hand | baseline in mTLSS | 3 (severe) to each component, giving a maximum disease severity of 21. The | missing, that domain is missing. |
| Scale | eczema (HE) lesion severity (erythema,<br>edema, desquamation, fissures,<br>hyperkeratosis or lichenification, and<br>vesicles) with the intensity of pruritus | | recall period for this scale is the present time. | |

| | or pain to assess the severity of symptoms. | | | |
|---|---|---|---|---|
| Pruritis<br>Numeric<br>Rating Scale<br>(NRS) | The Pruritus Numeric Rating Scale (NRS) is a participant-reported, single-item, daily, 11-point scale. | Percent change from baseline Pruritis NRS Score 4-point improvement in Pruritis NRS Score 3-point improvement in Pruritus NRS Score | The Pruritus NRS is used by participants to rate their worst itch severity over the past 24 hours with 0 indicating "No itch" and 10 indicating "Worst itch imaginable." Assessments will be recorded daily by the participant. The minimal clinically important change is 3 points. Participants will record the pruritus assessments daily using an electronic diary at home. As indicated in the SoA (Section 1.3), initial electronic diary entries for Pruritus NRS should be completed a minimum of 4 of 7 days before baseline. | Baseline weekly mean score is missing if the patient has 3 or fewer responses within the week before baseline. Post-baseline weekly mean score is missing if the patient has no responses within the week. |
| Skin Pain<br>Numeric<br>Rating Scale<br>(NRS) | The Skin Pain NRS is a participant-reported, 11-point horizontal scale anchored at 0 and 10, with 0 representing "no pain" and 10 representing "worst pain imaginable." | Percent change from<br>baseline in Skin Pain<br>NRS Score<br>4-point improvement in<br>Skin Pain NRS Score | Overall severity of a participant's skin pain is indicated by selecting the number that best describes the worst level of skin pain in the past 24 hours. Assessment will be recorded daily by the participant. | Baseline weekly mean score is missing if the patient has 3 or fewer responses within the week before baseline. Post-baseline weekly mean score is missing if the patient has no responses within the week. |
| Sleep-Loss<br>Scale | The Sleep-Loss Scale is a participant-reported, single-item, daily scale that measures the extent of sleep loss due to interference of itch over the last night. | Percent change from baseline in Sleep Loss Score 2-point improvement in Sleep Loss Score | The Sleep-Loss Scale is rated based on a 5-point Likert scale (0 [not at all] to 4 [unable to sleep at all]). Assessment will be recorded daily by the participant. The minimal clinically important change is 3 points. | Baseline weekly mean score is missing if the patient has 3 or fewer responses within the week before baseline. Post-baseline weekly mean score is missing if the patient has no responses within the week. |

| Atopic | The Atopic Dermatitis Control Tool is a | Percent change from | Each of the 6 Atopic Dermatitis Control | If 1 question in a domain is |
|---|---|---|---|---|
| Dermatitis | patient-reported, simple, brief tool for | baseline in ADCT Total | Tool items has a score range from 0 (no | missing, that domain is |
| Control Tool | adults and adolescents that evaluates 6 | Score | problem) to 4 (worst), rating the | missing. |
| | symptoms and effects associated with | | severity of each concept; the total score | 8 |
| | AD over the past week | | ranges from 0 to 24, which is the | |
| | 1 | | summation of the responses to all the | |
| | | | items. A score of ≥7 points was derived | |
| | | | as the threshold to identify participants | |
| | | | "not in control." The threshold for | |
| | | | meaningful within-person change was | |
| | | | estimated | |
| | | | to be 5 points. | |
| Participant | The question on participant satisfaction | PRSQ Score | The response options range from 1 (not | Single item, missing if |
| Reported | asks "How satisfied are you with this | | satisfied) to 5 (completely satisfied). | missing. |
| Satisfaction | treatment's ability to treat your skin | | | |
| Question | condition?" | | | |
| WPAI-AD | The Work Productivity and Activity | Percent change from | The Work Productivity and Activity | If 1 question in a domain is |
| | Impairment Questionnaire-Atopic | baseline in WPAI AD | Impairment Questionnaire- Atopic | missing, that domain is |
| | Dermatitis is a participant-reported, 6- | Absenteeism Score | Dermatitis consists of 6 items grouped | missing. |
| | item questionnaire that records | | into 4 domains: absenteeism (work time | |
| | impairment due to AD over the past 7 | Percent change from | missed), presenteeism (impairment at | |
| | days in adolescents and adults | baseline in WPAI AD | work or reduced on the job | |
| | | Presenteeism Score | effectiveness), work productivity loss | |
| | | | (overall work impairment or | |
| | | Percent change from | absenteeism plus presenteeism), and | |
| | | baseline in WPAI AD | activity impairment. Absenteeism, | |
| | | Work Productivity Loss | presentism, and work productivity will | |
| | | Score | only be reported by those who are | |
| | | D . 1 . C | currently employed (working for pay) at | |
| | | Percent change from | the time of the scale completion. The | |
| | | baseline in WPAI AD | recall period for the scale is | |
| | | Activity Impairment Score | over the past 7 days. Scores are | |
| | | Score | calculated as impairment percentages | |
| | | | (Reilly et al. 1993), with | |
| | | | higher scores indicating greater | |

| impairment and less productivity |
|----------------------------------|
| F |

Abbreviations: AD = atopic dermatitis; HRQoL = health-related quality of life; NA = not applicable; QoL = quality of life.

<sup>&</sup>lt;sup>a</sup> Secondary endpoints.

#### 5.12. Health Outcomes/Quality-of-Life Analyses

The description and derivation of the health outcomes/QoL analyses are described in Table KGBO.5.4. For categorical parameters, the number and percentage of patients in each category will be presented, as well as a 90% Wilson-Score confidence interval for the percentage. For continuous parameters, descriptive statistics will include n (number of patients), mean, standard deviation, Q1, median, Q3, minimum, and maximum. These summaries will be provided for the data as-observed and after implementation of LOCF and MCMC-MI imputation as described in Sections 5.4.2. and 5.4.3. Patient-Reported Outcomes Information System and DLQI/CDLQI will be reported by clinic visit.

#### 5.13. Safety Analyses

The planned analyses of safety data will be performed with an intent to maintain consistency with compound-level standard safety analyses. These standards are based on internal standards which were informed by CDISC standards, regulatory guidance (eg, FDA Clinical Review Template), and cross-industry standardization efforts (eg, PhUSE white papers from the Standard Analyses and Code Sharing Working Group provided in the PhUSE Computational Science Deliverables Catalog [WWW]).

The laboratory (including hormone), vital sign (including growth), and immunogenicity safety summaries will be based on the safety population. The extent of exposure and AE tables will be based on the safety population.

These analysis populations are fully defined in Table KGBO.5.1.

Not all displays described in this section will necessarily be included in the CSRs. Any display described and not provided in the CSR would be available upon request. Not all displays will necessarily be created as a "static" display. Some may be incorporated into interactive display tools instead of or in addition to a static display. Any display created interactively will be included in the CSR if deemed relevant to the discussion.

#### 5.13.1. Extent of Exposure

A by-patient listing of exposure duration with the number of active injections and total dose will be provided for the Safety Population.

The duration of exposure will be calculated as:

*Duration of exposure (days) =* 

Date of last visit (scheduled or unscheduled) in the Treatment Period –

*Date of first dose+1* 

The number and percentage of patients in each of the following categories will be included in the summaries:

 $>0, \ge 7$  days,  $\ge 14$  days,  $\ge 30$  days,  $\ge 60$  days,  $\ge 90$  days,  $\ge 112$  days,  $\ge 120$  days,  $\ge 168$  days. Note that patients may be included in more than 1 category.

The summaries will also include the following information:

• total exposure in patient years, calculated as:

Total exposure in patient years  $= \frac{Sum \ of \ duration \ of \ exposures \ for \ all \ patients \ in \ treatment \ group}{365.25}$ 

- mean and median total dose; total dose (in mg) is calculated by the number of active injections taken multiplied by 250.
- Total number of injections received will be derived from the *Exposure as Collected* eCRF page and on the *Exposure as Collected: Missed Injections at Home* eCRF page.

#### 5.13.2. Adverse Events

A TEAE is defined as an event that first occurred or worsened in severity after baseline (ie, AEs with an onset date on or after the date of the first injection of study drug). The MedDRA lowest-level term will be used in the treatment-emergent computation. The maximum severity for each lowest-level term during the baseline period will be used as baseline. The treatment period will be included as post-baseline for the summaries. For events with a missing severity during the baseline period, the events will be treated as 'mild' in severity for determining treatment-emergence. Events with a missing severity during the postbaseline period will be treated as 'severe', and treatment-emergence will be determined by comparing to baseline severity. For events occurring on the day of first taking study medication, the events will be assumed to be posttreatment.

The planned summaries for AEs are provided in Table KGBO.5.5 and are described more fully in compound-level safety standards and in the AE-related PhUSE white paper [Analysis and Displays Associated with Adverse Events: Focus on Adverse Events in Phase 2-4 Clinical Trials and Integrated Summary Document (PhUSE 2017)].

Summary tables will be presented for the safety population. Summary tables will include the number and percentage of patients reporting an event. For events that are gender-specific (as defined by MedDRA), the number of participants at risk will include only patients from the given gender.

Table KGBO.5.5.Summary Tables/Listings Related to Adverse Events

| Summaries | Population |
|---|---|
| Overview of AEs | Safety |
| Summary of TEAEs by PTs | Safety |
| Summary of TEAEs by PTs within SOC | Safety |
| Summary of TEAE PTs by maximum severity | Safety |
| Summary of SAEs by PT within SOC | Safety |
| Summary of AEs leading to treatment discontinuation by PT with SOC | Safety |

| Summary of TEAEs possibly related to study drug by PTs within SOC | Safety |
|---|---|
| Summary of treatment-emergent adverse events – facial dermatitis follow-up form | Safety |
| Listing of SAEs (including Death) | Safety |
| Listing of primary AEs leading to study treatment discontinuation | Safety |
| Listing of TEAEs | Safety |

Abbreviations: AE = adverse event; PT = Preferred Term; SAE = serious adverse event; SOC = System Organ Class; TEAE = treatment-emergent adverse event.

#### 5.13.2.1. Common Adverse Events

The percentages of patients with TEAEs will be summarized using MedDRA PT for the common TEAEs (occurred in  $\geq$ 1% before rounding in any column in the table).

## 5.13.2.2. Deaths, Other Serious Adverse Events and Other Notable Adverse Events

The number and percentage of patients reported with an SAE during the treatment period will be summarized using MedDRA PT. A listing of SAEs will be provided.

The number and percentage of patients who permanently discontinued from study treatment due to an AE (including AEs that led to death) during the treatment period will be summarized using MedDRA PT. Events will be ordered by decreasing frequency.

#### 5.13.3. Clinical Laboratory Evaluation

As described more fully in compound-level safety standards and in the laboratory-related PhUSE white papers (PhUSE 2013; PhUSE 2015), the clinical laboratory evaluations will be summarized as described in Table KGBO.5.6. Hormone analytes are summarized/plotted similarly.

Table KGBO.5.6.Summary Tables/Listing of Clinical Laboratory Evaluations

| Summaries | Population |
|---|---|
| Box plots of observed values by visit | Safety |
| Box plots for change from baseline values by visit | |
| Change from baseline to last observations | Safety |
| Treatment-emergent abnormal high lab values (ie, patients shifting from a normal/low maximum baseline value to a high maximum postbaseline value) or abnormal low lab values (ie, patients shifting from normal/high minimum baseline value to a low minimum postbaseline value) | Safety |
| Shift tables showing the number of patients who shift from each category of maximum (minimum) baseline observation to each category of maximum (minimum) postbaseline observation. Here categories may be low, normal, or high with cut-offs defined in the compound-level safety standards. | Safety |
| Listing of abnormal findings for laboratory analyte measurements, including qualitative measures | Safety |

#### 5.13.4. Vital Signs and Other Physical Findings

As described more fully in compound-level safety standards and in the laboratory-related PhUSE white papers (PhUSE 2013; PhUSE 2015), vital signs will be summarized similarly to the clinical laboratory evaluation (Table KGBO.5.7). For vital signs, treatment-emergent low and high are based on a combination of a specified value and a change or percentage change as defined in the compound-level safety standards.

Table KGBO.5.7. Summary Tables/Figures Related to Vital Signs

| Summaries | Population |
|---|---|
| Box plots for observed values by visit | Safety |
| Box plots for change from baseline values by visit | Safety |
| Tables with the number and percentage of subjects who shift from normal/high to low (ie, treatment-emergent low) and the number and percentage of subjects who shift from normal/low to high (ie, treatment-emergent high); the limits are defined in the compound-level safety standards | Safety |

#### 5.13.5. Immunogenicity

Anti-drug antibodies (ADA) analysis will only occur upon request from, for example, regulatory or a business need. An individual sample will be potentially examined multiple times in a hierarchical procedure to produce a sample ADAs assay result and may yield a sample NAb assay result. Treatment-emergent ADAs are defined as those with a titer 2-fold (1 dilution) greater than the minimum required dilution if no ADAs were detected at baseline (treatment-induced ADA) or those with a 4-fold (2 dilutions) increase in titer compared to baseline if ADAs were detected at baseline (treatment-boosted ADA). A patient is considered TE-ADA positive when at least 1 postbaseline ADA sample meets the definition of TE-ADA.

Compound-level safety standards will be followed in the analyses of immunogenicity. Listings of immunogenicity assessments will be provided along with the summary of specified TEAEs by

TE-ADA status. The summary of TE-ADA and NAb status will be produced for the Safety Population.

# 5.13.6. Special Safety Topics including Adverse Events of Special Interest

This section includes areas of interest whether due to observed safety findings, potential findings based on drug class, or safety topics anticipated to be requested by a regulatory agency for any reason. In general, potential AESI relevant to these special safety topics will be identified by 1 or more SMQs, by a Lilly-defined MedDRA PT listing based upon the review of the most current version of MedDRA, or by treatment-emergent relevant laboratory changes, as described below. Additional special safety topics may be added as warranted.

Unless otherwise specified, the AESI will be summarized for the safety population.

Full details of the search terms and rules for deriving AESI in each of the sections below are described in the compound-level safety standards along with information about the types of summaries and listings to be provided. In the event that the listing of terms or analysis changes for a special safety topic, it will be documented in the compound-level safety standards, which will supersede this document; it will not warrant an amendment to the individual study SAP.

#### 5.13.6.1. Hepatic Safety

Hepatic labs include alanine aminotransferase (ALT) aspartate transaminase (AST), total bilirubin (TBL), and serum alkaline phosphatase (ALP).

Table KGBO.5.8. Summary Tables/Figure Related to Hepatic Safety

| Summaries | Population |
|---|---|
| ALT and AST: The number and percentage of subjects with a measurement greater than | Safety |
| or equal to 3 times (3X), 5 times (5X), and 10 times (10X) the performing lab ULN | |
| during the treatment period for all subjects with a postbaseline value and for subsets | |
| based on various levels of baseline value | |
| TBL and ALP: The number and percentage of subjects with a measurement greater than | |
| or equal to 2 times (2X) the performing lab ULN during the treatment period will be | |
| summarized for all subjects with a postbaseline value and for subsets based on various | |
| levels of baseline value | |
| Plot of maximum postbaseline ALT vs. maximum postbaseline total bilirubin | Safety |

Abbreviations: ALP = serum alkaline phosphatase; ALT = alanine aminotransferase; AST = aspartate transaminase; TBL = total bilirubin; ULN = upper limit of normal.

#### 5.13.6.2. Eosinophilia and Eosinophil-Related Disorders

In addition to the standard laboratory summaries (Section 5.13.3), eosinophilia and eosinophil-related AEs will be summarized. Details regarding- eosinophil-related PTs are in the compound-level safety standards.

Table KGBO.5.9. Summary Tables Related to Eosinophilia and Eosinophil-Related Adverse Events

| Summaries | Population |
|---|---|
| Shift table summarizing the number and percentage of participants within each | Safety |
| maximum baseline category versus each maximum postbaseline category | |

| Summary of eosinophil-related TEAE by PT Safety |
|-------------------------------------------------|
|-------------------------------------------------|

Abbreviations: AE = adverse event; PT = Preferred Term; TEAE = treatment-emergent adverse event.

# **5.13.6.3.** Infections, including herpes infections and relevant parasitic infections Infections will be defined using the PTs from the MedDRA Infections and Infestations SOC. The MedDRA terms used to identify infections considered to be opportunistic infections (OI) in patients with immune-mediated inflammatory conditions treated with immunomodulatory drugs are based on Winthrop et al. (2015) and are listed in the compound-level safety standards. The list contains narrow (more specific) and broad (less specific) PTs with respect to these prospectively defined OIs. Definitions of herpes infections, parasitic infections, and skin infections are listed in the compound-level safety standards.

Table KGBO.5.10. Summary Tables/Listing Related to Infection Related Adverse Events

| Summaries | Population |
|---|---|
| Summary of treatment-emergent infections by maximum severity | Safety |
| Summary of serious infections by PT | Safety |
| Summary of infection AEs resulting in permanent study drug discontinuation | Safety |
| Treatment-emergent adverse events - opportunistic and potential opportunistic infections | Safety |
| Treatment-emergent adverse events - herpes and parasitic infections | Safety |
| Treatment-emergent adverse events - skin infections | Safety |
| Treatment-emergent adverse events - infections characterization and follow-up form | Safety |
| Listing of patients with potential OIs, serious infections, herpes, and parasitic infections | Safety |

Abbreviations: AE = adverse event; OI = opportunistic infections; PT = Preferred Term.

#### 5.13.6.4. Conjunctivitis

Conjunctivitis events are events of special interest and will be identified using PTs nested within the categories of conjunctivitis and keratitis as described in the compound-level safety standards:

Table KGBO.5.11. Summary Table/Listing Related to Conjunctivitis

| Summaries | Population |
|---|---|
| Summary of TEAE of conjunctivitis and keratitis clusters | Safety |
| Treatment-emergent adverse events - conjunctivitis and eye inflammation | Safety |
| characterization follow-up form | |
| Listing of patients with conjunctivitis | Safety |

Abbreviation: TEAE = treatment-emergent adverse event.

#### 5.13.6.5. Hypersensitivity

Potential hypersensitivity reactions will be determined using the following SMQs: anaphylactic reaction, hypersensitivity, and angioedema. Potential hypersensitivity will be categorized as immediate (ie, occurring the same day as drug administration) and non-immediate (ie, occurring after the day of study drug administration but prior to subsequent drug administration). The planned summaries are provided in Table KGBO.5.12.

#### Table KGBO.5.12. Summary Tables/Listing Related to Hypersensitivity

| Summaries | Population |
|---|---|
| Treatment-emergent adverse events - potential immediate hypersensitivity reactions (events occurring on day of study drug administration) | Safety |
| Treatment-emergent adverse events - potential nonimmediate hypersensitivity reactions | Safety |
| (events occurring after day of study drug administration) | |

#### 5.13.6.6. Injection Site Reactions (ISRs)

Injection site reactions are AEs localized to the immediate site of the administration of a drug. The evaluation of study drug related ISRs will be through the unsolicited reporting of ISR TEAEs. Injection site reactions will be defined using the MedDRA high-level term (HLT) of ISR, excluding certain PTs (eg, those PTs related to injections into a joint) and administration site reactions as described in the compound-level safety standards.

Table KGBO.5.13. Summary Tables Related to Injection Site Reactions

| Summary | Population |
|-------------------------------------------|------------|
| Summary of TEAE of ISR overall, and by PT | Safety |

Abbreviations: HLT = high-level term; ISR = injection site reaction; PT = Preferred Term; TEAE = treatment-emergent adverse event.

#### 5.13.6.7. Malignancies

Malignancies will be defined using PTs from the Malignant tumors SMQ and summarized separately for the 2 categories: Non-melanoma skin cancer (NMSC) and malignancies excluding NMSC.

Table KGBO.5.14. Summary Tables Related to Malignancies

| Summary | Population |
|---|---|
| Summary of TEAE of malignancies within categories of NMSC and malignancy | Safety |
| excluding NMSC | |

Abbreviations: NMSC = non-melanoma skin cancer; TEAE = treatment-emergent adverse event.

#### 5.13.6.8. Atopic Dermatitis Exacerbation

Atopic dermatitis exacerbation will be defined using PTs specified in the Compound Level Safety Standards and summarized for the Safety Population.

Table KGBO.5.15. Summary Tables Related to Atopic Dermatitis Exacerbation

| Analysis | Population |
|---------------------------------------------------|------------|
| Summary of TEAE of atopic dermatitis exacerbation | Safety |

Abbreviations: TEAE = treatment-emergent adverse event.

#### 5.13.6.9. Suicide/Self-Injury

The PTs from the suicide/self-injury SMO [20000037] will be summarized.

#### Table KGBO.5.16. Summary Tables Related to Suicidal Ideation and Behavior

| Analysis | Population |
|----------------------------------------|------------|
| Summary of TEAE of suicide/self-injury | Safety |

Abbreviations: TEAE = treatment-emergent adverse event.

#### 5.14. Subgroup Analyses

Subgroup analyses will be conducted for the primary endpoint, EASI-75 at Week 16, using descriptive statistics.

The following subgroups will be analyzed:

- weight category (<60 kg,  $\ge 60 \text{ to } <100 \text{ kg}$ , or  $\ge 100 \text{ kg}$ ).
- Age (12 to <18, 18+)
- Dupilumab Treatment Response (No response, Partial response, Lost Response)

Some additional subgroup analyses may be added. The analysis of additional subgroups will not require an amendment to the SAP.

#### 5.15. Protocol Deviations

Protocol deviations will be identified throughout the study. Important protocol deviations are defined as those deviations from the protocol likely to have a significant impact on the completeness, accuracy, and/or reliability of the study data or that may significantly affect a patient's rights, safety, or well-being.

Potential examples of important protocol deviations include patients who violated the inclusion/exclusion criteria, used an interfering concomitant medication, and significant non-compliance with study medication (<75% of expected injections). Refer to a separate document called "KGBO Trial Issues Management Plan" for the important protocol deviations with categorizations.

The number and percentage of patients having important protocol deviations will be summarized within category and subcategory of deviation for Weeks 0-16 of the Treatment Period using the ITT population and for Weeks 16-24 of the Treatment Period using the Treatment Period II Population.

A by-patient listing of important protocol deviations will be provided for the ITT population.

#### 5.16. Interim Analyses and Data Monitoring

Interim Analysis:

One interim analysis (primary lock) will be conducted after all enrolled participants have been evaluated at Week 16 or discontinued prior to Week 16. This interim database lock will include all efficacy and safety data collected by the cutoff date. Due to the open-label and descriptive nature of this study, there is no unblinding nor alpha adjustment.

Additional analyses and snapshots of study data may be performed to fulfill the need for regulatory interactions or publication purposes.

<u>Final DBL</u>: A final DBL will occur after all patients have either completed the study through the 12-week safety follow-up period of the study or discontinued the current study.

#### 5.17. Annual Report Analyses

Based on regulatory requirements for the DSUR, reports will be produced (if not already available from the study CSR) for the reporting period covered by the DSUR.

#### 5.18. Clinical Trial Registry Analyses

Additional analyses will be performed (if not already available from the study CSR) for the purpose of fulfilling the CTR requirements.

Analyses provided for the CTR requirements include the following:

Summary of AEs, provided as a dataset, will be converted to an XML file. Both SAEs and 'other' AEs are summarized by MedDRA PT.

- An AE is considered 'serious' whether or not it is a TEAE.
- An AE is considered in the 'other' category if it is both a TEAE and is not serious. For each SAE and 'other' AE, for each term the following are provided:
  - o the number of participants at risk of an event
  - o the number of participants who experienced each event term, and
  - o the number of events experienced.
- Consistent with www.ClinicalTrials.gov requirements, 'other' AEs that occur in <5% of patients/subjects may not be included if a 5% threshold is chosen (5% is the minimum threshold).
- AE reporting is consistent with other document disclosures (eg, the CSR, manuscripts, and so forth).

#### 5.19. Biomarker Analysis

Serum samples will be collected to discern responder variability within the study and to track response variability to lebrikizumab. Biomarkers will include but are not limited to:





Samples will be collected according to the schedule described in the SoA and as detailed in the laboratory manual provided separately to sites.

### 6. Unblinding Plan

Not applicable.

#### 7. References

- Auriemma M, Vianale G, Amerio P, Reale M. Cytokines and T cells in atopic dermatitis. Eur Cytokine Netw. 2013;24(1):37-44. https://doi.org/10.1684/ecn.2013.0333
- Basra MK, Salek MS, Camilleri L, et al. Determining the minimal clinically important difference and responsiveness of the Dermatology Life Quality Index (DLQI): further data. Dermatology. 2015;230(1):27-33. https://doi.org/10.1159/000365390
- Bieber T. Atopic dermatitis. N Engl J Med. 2008;358(14):1483-1494. https://doi.org/10.1056/nejmra074081
- Bieber T, Novak N. Pathogenesis of atopic dermatitis: new developments. Curr Allergy Asthma Rep. 2009;9(4):291-294. https://doi.org/10.1007/s11882-009-0041-2
- Bieber T. Atopic dermatitis 2.0: from the clinical phenotype to the molecular taxonomy and stratified medicine. Allergy. 2012;67(12):1475-1482. https://doi.org/10.1111/all.12049
- Bieber T. Interleukin-13: Targeting an underestimated cytokine in atopic dermatitis. Allergy. 2020;75(1):54-62. <a href="https://doi.org/10.1111/all.13954">https://doi.org/10.1111/all.13954</a>
- Bieber T, Straeter B. Off-label prescriptions for atopic dermatitis in Europe. Eur J Aller Clin Immunol. 2015;70(1):6-11. https://doi.org/10.1111/all.12498
- Bissonnette R, Diepgen T, Elsner P. Redefining treatment options in chronic hand eczema (CHE). J Eur Acad Dermatol Venereol. 2010;24(s3):1-20. https://doi.org/10.1111/j.14683083.2010.03615.x
- Caretti KL, Mehregan DR, Mehregan DA. A survey of self-reported skin disease in the elderly African-American population. Int J Dermatol. 2014;54(9):1034-1038. https://doi.org/10.1111/jjd.12520
- Choy DF, Hsu DK, Seshasayee D, et al. Comparative transcriptomic analyses of atopic dermatitis and psoriasis reveal shared neutrophilic inflammation. J Allergy Clin Immunol. 2012;130(6):1335-1343. <a href="https://doi.org/10.1016/j.jaci.2012.06.044">https://doi.org/10.1016/j.jaci.2012.06.044</a>
- Diepgen T, Ofenloch R, Bruze M, et al. Prevalence of contact allergy in the general population in different European regions. British J Dermatol. 2016;174:319-329. https://doi.org/10.1111/bjd.14167
- Eckert L, Gupta S, Amand C, et al. The burden of atopic dermatitis in US adults: Health care resource utilization data from the 2013 National Health and Wellness Survey. J Am Acad Dermatol. 2018;78(1):54-61.e1. https://doi.org/10.1016/j.jaad.2017.08.002
- Eckert L, Gupta S, Gadkari A, et al. Burden of illness in adults with atopic dermatitis: Analysis of National Health and Wellness Survey data from France, Germany, Italy, Spain, and the United Kingdom. J Am Acad Dermatol. 2019;81(1):187-195. https://doi.org/10.1016/j.jaad.2019.03.037
- Esche C, de Benedetto A, Beck LA. Keratinocytes in atopic dermatitis: inflammatory signals. Curr Allergy Asthma Rep. 2004;4(4):276-284. https://doi.org/10.1007/s11882-004-0071-8

Faiz S, Giovannelli J, Podevin C et al. Effectiveness and safety of dupilumab for the treatment of atopic dermatitis in a real-life French multicenter adult cohort. J Am Acad Dermatol. 2019;81:143-51. https://doi.org/10.1016/j.jaad.2019.02.053

Faiz S, Giovannelli J, Podevin C et al. Effectiveness and safety of dupilumab for the treatment of atopic dermatitis in a real-life French multicenter adult cohort. J Am Acad Dermatol. 2019

Gooderham MJ, Hong HC, Eshtiaghi P, Papp KA. Dupilumab: A review of its use in the treatment of atopic dermatitis. Am Acad Dermatol. 2018;78(3):S28-S36. https://doi.org/10.1016/j.jaad.2017.12.022

Hamid Q, Naseer T, Minshall EM, et al. In vivo expression of IL-12 and IL-13 in atopic dermatitis. J Allergy Clin Immunol. 1996;98(1):225-231. https://doi.org/10.1016/s00916749(96)70246-4

Hanifin JM, Thurston M, Omoto M, et al. EASI Evaluator Group. The eczema area and severity index (EASI): assessment of reliability in atopic dermatitis. Exp Dermatol. 2001;10(1):11-18. https://doi.org/10.1034/j.1600-0625.2001.100102.x

Harrop J, Chinn S, Verlato G, et al. Eczema, atopy and allergen exposure in adults: a population based study. Clin Exper Aller. 2007;37:526-535. https://doi.org/10.1111/j.13652222.2007.02679.x

He JQ, Chan-Yeung M, Becker AB, et al. Genetic variants of the IL13 and IL4 genes and atopic diseases in at-risk children. Genes Immun. 2003;4(5):385-389.

Heibel H, Henddricks A, Foshee J, Shi V. Rosacea associated with dupilumab therapy. J Dermatol Treat. 2021;32(1):114-116. https://doi.org/10.1080/09546634.2019.1624683

High WA, Tomasini CF, Argenziano G, Zalaudek I. Basic principles of dermatology. In: Bolognia JL, Jorizzo JL, Schaffer JV, editors. Dermatology (3rd ed.). China: Elsevier; 2012: pp. 8

Hongbo Y, Thomas CL, Harrison MA, et al. Translating the science of quality of life into practice: What do dermatology life quality index scores mean? J Invest Dermatol. 2005;125(4):659-664. https://doi.org/10.1111/j.0022-202x.2005.23621.x

Howell MD, Fairchild HR, Kim BE, et al. Th2 cytokines act on S100/A11 to downregulate keratinocyte differentiation. J Invest Dermatol. 2008;128(9):2248-2258. https://doi.org/10.1038/jid.2008.74

Hua TC, Hwang CY, Chen YJ, et al. The natural course of early-onset atopic dermatitis in Taiwan: a population-based cohort study. Br J Dermatol. 2014;170(1):130-135. https://doi.org/10.1111/bjd.12603

Hummelshoj T, Bodtger U, Datta P, et al. Association between an interleukin-13 promoter polymorphism and atopy. Eur J Immunogenet. 2003;30(5):355-359. https://doi.org/10.1046/j.1365-2370.2003.00416.x Illi S, von Mutius E, Lau S, et al. The natural course of atopic dermatitis from birth to age 7 years and the association with asthma. J Allergy Clin Immunol. 2004;113(5):925-931. https://doi.org/10.1016/j.jaci.2004.01.778

Jeong CW, Ahn KS, Rho NK, et al. Differential in vivo cytokine mRNA expression in lesional skin of intrinsic vs. extrinsic atopic dermatitis patients using semiquantitative RT-PCR. Clin Exp Allergy. 2003;33(12):1717-1724. https://doi.org/10.1111/j.1365-2222.2003.01782.x

Kiebert, G, Sorensen SV, Revicki D, et al. Atopic dermatitis is associated with a decrement in health-related quality of life. Int J Dermatol. 2002;41(3):151-158. <a href="https://doi.org/10.1046/j.1365-4362.2002.01436.x">https://doi.org/10.1046/j.1365-4362.2002.01436.x</a>

Kim BE, Leung DYM, Boguniewicz M, Howell MD. Loricrin and involucrin expression is down-regulated by Th2 cytokines through STAT-6. Clin Immunol. 2008;126(3):332-337. <a href="https://doi.org/10.1016/j.clim.2007.11.006">https://doi.org/10.1016/j.clim.2007.11.006</a>

Khilji FA, Gonzalez M, Finlay AY. Clinical meaning of change in Dermatology Life Quality Index scores. Br J Dermatol. 2002;147:25-54.

Kunz B, Oranje AP, Labrèze L, et al. Clinical validation and guidelines for the SCORAD index: consensus report of the European Task Force on Atopic Dermatitis. Dermatology. 1997;195(1):10-19. https://doi.org/10.1159/000245677

La Grutta S, Richiusa P, Pizzolanti G, et al. CD4(+)IL-13(+) cells in peripheral blood well correlates with the severity of atopic dermatitis in children. Allergy. 2005;60(3):391-395. https://doi.org/10.1111/j.1398-9995.2005.00733.x

Langan SM, Irvine AD, Weidinger S. Atopic dermatitis. Lancet. 2020;396(10247):345-360. https://doi.org/10.1016/s0140-6736(20)31286-1

Marniquet M, Seneschal J, Darrigade A, et al. Reasons for discontinuation of dupilumab in adult atopic dermatitis in clinical practice. Br J Dermatol. 2022. https://doi.org/10.1111/bjd.20883

Miron Y, Miller P, Hughes C, et al. Mechanistic insights into the antipruritic effects of lebrikizumab, an anti–IL-13 mAb. J Aller Clin Immun. 2022. 1-11. https://doi.org/10.1016/j.jaci.2022.01.028

Neis MM, Peters B, Dreuw A, et al. Enhanced expression levels of IL-31 correlate with IL-4 and IL-13 in atopic and allergic contact dermatitis. J Allergy Clin Immunol. 2006;118(4):930-937. https://doi.org/10.1016/j.jaci.2006.07.015

Newton L, DeLozier AM, Griffiths PC, et al. Exploring content and psychometric validity of newly developed assessment tools for itch and skin pain in atopic dermatitis. J Patient Rep Outcomes. 2019;3(1):42. <a href="https://doi.org/10.1186/s41687-019-0128-z">https://doi.org/10.1186/s41687-019-0128-z</a>

Novak N, Kruse S, Kraft S, et al. Dichotomic nature of atopic dermatitis reflected by combined analysis of monocyte immunophenotyping and single nucleotide polymorphisms of the interleukin-4/interleukin-13 receptor gene: the dichotomy of extrinsic and intrinsic atopic

dermatitis. J Invest Dermatol. 2002;119(4):870-875. https://doi.org/10.1046/j.15231747.2002.00191.x

Oranje AP, Glazenburg EJ, Wolkerstorfer A, de Waard-van der Spek FB. Practical issues on interpretation of scoring atopic dermatitis: the SCORAD index, objective SCORAD and the three-item severity score. Br J Dermatol. 2007;157(4):645-648. https://doi.org/10.1111/j.13652133.2007.08112.x

Pariser DM, Simpson EL, Gadkari A, et al. Evaluating patient-perceived control of atopic dermatitis: design, validation, and scoring of the Atopic Dermatitis Control Tool (ADCT). Curr Med Res Opin. 2020;36(3):367-376. <a href="https://doi.org/10.1080/03007995.2019.1699516">https://doi.org/10.1080/03007995.2019.1699516</a>

Purwar R, Werfel T, Wittmann M. IL-13-stimulated human keratinocytes preferentially attract CD4+CCR4+ T cells: possible role in atopic dermatitis. J Invest Dermatol. 2006;126(5):1043-1051. https://doi.org/10.1038/sj.jid.5700085

Reilly MC, Zbrozek AS, Dukes EM. The validity and reproducibility of a work productivity and activity impairment instrument. Pharmacoeconomics. 1993;4(5):353-365. https://doi.org/10.2165/00019053-199304050-00006

Ruzicka T, Harsch M, Brown TC, et al. Modified Total Lesion Symptom Score (mTLSS). Br J Dermatol. 2008;158(4):808-817.

Sacotte R, Silverberg J. Epidemiology of adult atopic dermatitis. Clin Dermatology. 2018;36:595-605. <a href="https://doi.org/10.1016/j.clindermatol.2018.05.007">https://doi.org/10.1016/j.clindermatol.2018.05.007</a>

Saeki H, Tsunemi Y, Fujita H, et al. Prevalence of atopic dermatitis determined by clinical examination in Japanese adults. J Dermatol. 2006;33(11):817-819. https://doi.org/10.1111/j.1346-8138.2006.00187.x

Safa G, Paumier V. Psoriasis induced by dupilumab therapy. Clin Exp Dermatol. 2019;44(3):e49-e50. https://doi.org/10.1111/ced.13901

Schram ME, Spuls PI, Leeflang MMG, et al. EASI, (objective) SCORAD and POEM for atopic eczema: responsiveness and minimal clinically important difference. Allergy. 2012;67(1):99106. <a href="https://doi.org/10.1111/j.1398-9995.2011.02719.x">https://doi.org/10.1111/j.1398-9995.2011.02719.x</a>

Seegräber M, Srour J, Walter A, et al. Dupilumab for treatment of atopic dermatitis. Expert Rev Clin Pharmacol. 2018;11(5):467-474. https://doi.org/10.1080/17512433.2018.1449642

Silverberg JI, Gelfand JM, Margolis DJ, et al. Patient burden and quality of life in atopic dermatitis in US adults: A population-based cross-sectional study. Ann Allergy, Asthma Immunol. 2018;121(3):340-347. <a href="https://doi.org/10.1016/j.anai.2018.07.006">https://doi.org/10.1016/j.anai.2018.07.006</a>

Silverberg JI. Comorbidities and the impact of atopic dermatitis. Ann Allergy, Asthma Immunol. 2019;123(2):144-151. https://doi.org/10.1016/j.anai.2019.04.020

Silverberg JI, DeLozier A, Sun L, et al. Psychometric properties of the itch numeric rating scale, skin pain numeric rating scale, and atopic dermatitis sleep scale in adult patients with

moderateto-severe atopic dermatitis. Health Qual Life Outcomes. 2021;19(1):247. <a href="https://doi.org/10.1186/s12955-021-01877-8">https://doi.org/10.1186/s12955-021-01877-8</a>

Simon D, Wollenberg A, Renz H, Simon HU. Atopic dermatitis: Collegium Internationale Allergologicum (CIA) update 2019. Int Arch Allergy Immunol. 2019;178(3):207-218. https://doi.org/10.1159/000497383

Simpson E, Bieber T, Guttman-Yassky E, et al. Two phase 3 trials of dupilumab versus placebo in atopic dermatitis. N Engl J Med. 2016;375:2335-2348. https://doi.org/10.1056/nejmoa1610020

#### **Appendix 1.** Definition of Rescue Medications

The AD rescue therapy in this study is defined as: high-potency TCS >10 days, topical JAK inhibitors (i.e. topical Ruxolitinib), and systemic AD therapy. The topical and systemic treatments are defined as follows:

#### 1. Topical AD Treatment (including TCSs, TCI, crisaborole, and Ruxolitinib)

Route of topical treatments includes: Topical and Transdermal.

TCS: ATC code is D07

High Potency TCS: ATC codes are D07AC or D07AD

Low or moderate potency TCS: ATC code is D07, excluding D07AC or D07AD

TCI: PT includes: TACROLIMUS, PIMECROLIMUS

Crisaborole: PT includes: CRISABOROLE

Topical Ruxolitinib: ATC code is D11AH09

## 2. Systemic AD Treatment (including systemic corticosteroids, immunosuppressant, biologics, and phototherapy/PUVA)

Route of systemic treatments administration includes: Oral, Intra-Arterial, Intramuscular, Intraperitoneal, Intravenous, Subcutaneous, and Transdermal. (This condition applies to the following categories except for phototherapies.)

Systemic Corticosteroids: ATC code is H02

<u>Immunosuppressant</u>: Defined as: ATC2 is L04 or PTs of Abrocitinib or Ruxolitinib excluding PTs mentioned in Biologics

Biologics: Defined as following PTs:

Infliximab, Infliximabum, Etanercept, Etanerceptum, Adalimumab, Adalimumabum, Certolizumab, Certolizumabum, Certolizumab pegol, Golimumab, Golimumabum, Ozoralizumab, Afelimomab, Afelimomabum, Tumor Necrosis Factor Alpha (TNF-) Inhibitors, Tabalumab, Tregalizumab, Anakinra, Basiliximab, Basiliximabum, Daclizumab, Daclizumabum, Tocilizumab, Tocilizumabum, Mepolizumab, Mepolizumab, Mepolizumabum, Rilonacept, Rilonaceptum, Ustekinumab, Canakinumab, Briakinumab, Fezakinumab, Sirukumab, Sarilumab, Lebrikizumab, Secukinumab, Olokizumab, Gevokizumab, Brodalumab, Ladarixin, Ixekizumab, Dupilumab, Tildrakizumab, Tildrakizumab, Reslizumabum, Guselkumab, Guselkumabum, Olamkicept, Fletikumab, Bimekizumab, Mirikizumab, Risankizumab, Abatacept, Ligelizumab, Vedolizumab, Belimumab, Nemolizumab, Tralokinumab, Omalizumab

#### **Phototherapy or PUVA:**

Programming search of medication name (actual term or PT) contains 'photo' then medicals to manually review to confirm whether the medication in question is indeed 'Phototherapy' or 'Photochemotherapy'.

